CLINICAL TRIAL: NCT01934192
Title: NUTRItional Adequacy Therapeutic Enhancement in the Critically Ill: A Randomized Double Blind, Placebo-controlled Trial of the Motilin Receptor Agonist GSK962040. The NUTRIATE Study
Brief Title: Nutritional Adequacy Therapeutic Enhancement in the Critically Ill. The NUTRIATE Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113445
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-10

CONDITIONS: Gastroparesis
Keywords: tolerability; camicinal; single dose; acetaminophen; gastric emptying; critically ill; GSK962040; pharmacokinetics; pharmacodynamics; gut motility
MeSH Terms: conditions — Gastroparesis; Critical Illness | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Initial randomization: GSK962040 Arm (Experimental): Subjects in the GSK962040 Arm will receive 50 mg once daily enteral dose administered through NG tube up to 7 days.
  Interventions: Drug: GSK962040 50 mg
- Initial randomization: Placebo Arm (Placebo Comparator): Subjects in the placebo arm will receive once daily dose enteral dose administered through NG tube up to 7 days.
  Interventions: Drug: Placebo NG
- Treatment change due to intolerance: GSK962040 Arm (Experimental): Subjects that develop intolerance and that originally received Placebo will receive 50 mg once daily enteral dose administered through NG tube + placebo IV
  Interventions: Drug: GSK962040 50 mg; Drug: Placebo IV
- Treatment change due to intolerance: Metoclopramide Arm (Active Comparator): Subjects that develop intolerance and that originally received GSK962040 will receive metoclopramide 10 mg IV every 6 h + placebo NG
  Interventions: Drug: Metoclopramide 10 mg; Drug: Placebo NG

INTERVENTIONS:
Drug: GSK962040 50 mg — GSK962040 50 mg will be administered once daily enteral dose through NG tube up to 7 days.
  Arms: Initial randomization: GSK962040 Arm; Treatment change due to intolerance: GSK962040 Arm
Drug: Metoclopramide 10 mg — Metoclopramide will be administered IV every 6 h
  Arms: Treatment change due to intolerance: Metoclopramide Arm
Drug: Placebo NG — Matching placebo once daily enteral dose will be administered through NG tube up to 7 days
  Arms: Initial randomization: Placebo Arm; Treatment change due to intolerance: Metoclopramide Arm
Drug: Placebo IV — Placebo will be administered IV every 6 hours
  Arms: Treatment change due to intolerance: GSK962040 Arm

SUMMARY:
This is a multi-center, parallel group, placebo-controlled and active-compared, randomized study to assess the ability of GSK962040 to enhance the delivery of enteral feed to critically ill subjects that are predisposed to developing feeding intolerance (e.g., percentage of goal volume); enhance gastric emptying in this population; and provide preliminary evidence of the drug's effect on outcomes of therapy (length of stay in the Intensive Care Unit [ICU], time on ventilator, ICU acquired infections, and 60-day mortality). Other aims are evaluation of GSK962040 safety, tolerability and pharmacokinetics upon repeat dosing in a critically ill population.

After meeting eligibility criteria, male and female subjects will be randomized to either receive GSK962040 (50 milligram [mg]) once daily (OD) via naso-gastric (NG) or orogastric (OG) feeding tube (oral solution), or placebo by the same route. If subjects develop intolerance to enteral feeding at any point up to Dose 5 of study medication (inclusive), study treatments will switch such that those originally receiving GSK962040 will receive metoclopramide (10 mg, intravenous [iv], every 6 hours) and those subjects originally randomized to receive placebo will receive GSK962040 (50 mg, via NG, OD). Additionally, if subjects develop intolerance prior to any treatment, they will be randomized to receive either GSK962040 (50 mg, via NG, OD) or metoclopramide (10 mg, iv, every 6 hours).

The study will consist of a screening/baseline assessment, a treatment period (up to 7 days in duration), and a 4-day post treatment safety follow-up assessment. The duration of each subject's participation in the study from screening to follow-up safety assessment will be up to approximately 2 weeks. In addition, mortality will be assessed 60 days after admission to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age & Gender: Male or female between 18 and 85 years of age inclusive, at the time of obtaining the informed consent.
* First admitted to participating ICU within the previous 48 hours.
* Intubated and invasively mechanically ventilated
* Indicated to receive early EN or are already receiving EN (subject must be on EN prior to receiving study treatment)
* Have at least one of the following
* Clinical evidence of cardiovascular dysfunction defined as the need for vasopressor agents (e.g. norepinephrine, epinephrine, vasopressin), >5 microgram/kg/min of dopamine, or >/= 50 microgram/min phenylephrine) for greater than or equal to 2 hours;
* Poly-trauma with an injury severity score (ISS) >=15 points
* Acute traumatic or non-traumatic brain injury Glasgow Coma Scale (GCS) <=12, prior to the initiation of sedation.

Exclusion Criteria:

* Subjects who are not expected to be in the ICU and alive for at least 48 hrs from point of screening.
* Subjects with acute hepatitis (e.g. acute hepatitis B or C) or severe chronic liver disease (e.g. Child Pugh class C cirrhosis) will be excluded
* Liver function tests: If Alanine aminotransferase (ALT) >=8x upper limit of normal (ULN); OR If ALT >5-8x ULN and bilirubin >2<=3 ULN or bilirubin >3x ULN (Include only if bilirubin <1.5xULN); OR If ALT <=5xULN and Bilirubin >3xULN (Include only if ALT <=3xULN and Bilirubin >2 <=3xULN)
* Subjects who have received a gastric prokinetic agent in the previous 12 hours (e.g., erythromycin, azithromycin, metoclopramide, domperidone).
* QT duration corrected for heart rate (QTc) >480 ms. QTcF is the recommended correction factor for all sites. If QT duration corrected for heart rate by Fridericia's formula (QTcF) is not possible to obtain or calculate, QT duration corrected for heart rate by Bazett's formula (QTcB) or machine or manual over read, may be obtained after consultation with the medical monitor. The QT correction formula used to determine inclusion and discontinuation should be the same throughout the study.
* Use of strong Cyp3A4 inhibitors
* Subjects who require renal replacement therapy or with an estimated glomerular filtration rate (GFR) of <30 mL/min byCockroft-Gault calculation).
* Subjects who have a history of or who have undergone major esophageal or gastric surgery on this admission (major lower abdominal surgery will not result in exclusion unless this carries a contraindication to enteral feeding).
* Subjects with an absolute contraindication to enteral nutrition e.g. subjects with ongoing bowel obstruction or perforation.
* Subject has a gastric pacemaker
* Pregnant or lactating females
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Concurrent enrollment in other interventional study involving a novel (i.e.unapproved or experimental) chemical or biopharmaceutical entity.
* Previous randomization in this study
* Subjects for whom the reason for admission to ICU was an overdose (deliberate or accidental; medicinal product or not).
* Exclusion to re-randomization:
* Subjects with an untreated pheochromocytoma.
* Subjects with a past history of a seizure disorder (e.g., epilepsy) and is currently receiving anti-epileptic treatment for their seizure disorder, ongoing refractory, or sustained seizure disorder (prophylactic use for head injury/isolated new seizure maintained on anti-seizure meds in ICU acceptable).
* Subjects taking drugs likely to cause extrapyramidal reactions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (4):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Philadelphia, Pennsylvania
- Australia (4):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Southport, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Woodville, South Australia
- Canada (9):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 92 participants between 18 to 85 years of age who were admitted to Intensive Care Unit (ICU), mechanically ventilated and who received enteral nutrition (EN) were included in this study.
Pre-assignment Details: The study consisted of a screening phase, a treatment period of up to 7 days and a post treatment safety follow-up of 14 days after the last dose of study medication. After performing Baseline tests eligible participants were included in the study.
Groups:
- Baseline EN Tolerant: Placebo/Camicinal: Participants who were tolerant to EN feeding at Baseline were randomized to receive up to 7 doses of placebo drug once daily via Naso-orogastric (NG) tube. Participants who developed intolerance to EN feeding at any point up to dose 5 were switched to receive Camicinal 50 milligram (mg) once daily along with placebo drug every 6 hours (hrs) via Intravenous (IV) route.
- Baseline EN Tolerant: Camicinal/Metoclopramide: Participants who were tolerant to EN feeding at Baseline were randomized to receive up to 7 doses of Camicinal (GSK962040) 50 mg once daily via NG tube. Participants who developed intolerance to EN feeding at any point up to dose 5 were switched to receive Metoclopramide 10 mg every 6 hrs via IV route along with placebo drug every 6 hrs via NG route.
- Baseline EN Intolerant: Camicinal: Participants who were intolerant to EN feeding at Baseline were randomized to receive Camicinal (GSK962040) 50 mg once daily via NG tube along with placebo drug every 6 hrs via IV route.
- Baseline EN Intolerant: Metoclopramide: Participant who were intolerant to EN feeding at Baseline were randomized to receive metoclopramide 10 mg every 6 Hrs. via IV route along with placebo drug every 6 hrs via NG tube.
Period: Overall Study
Arm/Group | Baseline EN Tolerant: Placebo/Camicinal | Baseline EN Tolerant: Camicinal/Metoclopramide | Baseline EN Intolerant: Camicinal | Baseline EN Intolerant: Metoclopramide
Started | 40 | 44 | 4 | 4
Completed | 31 | 37 | 3 | 3
Not Completed | 9 | 7 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Other: reached stopping criteria | 6 | 5 | 1 | 0
Not completed — Physician Decision | 3 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline EN Tolerant: Placebo/Camicinal | Baseline EN Tolerant: Camicinal/Metoclopramide | Baseline EN Intolerant: Camicinal | Baseline EN Intolerant: Metoclopramide | Total
Number analyzed (Participants) | 40 | 44 | 4 | 4 | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (15.93) | 59.8 (16.64) | 64.3 (13.40) | 45.5 (9.68) | 57.3 (16.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 2 | 1 | 27
  Male | 28 | 32 | 2 | 3 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Customized: American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Race, Customized: Asian - South East Asian Heritage | 0 | 1 | 0 | 0 | 1
  Race, Customized: White - White/Caucasian/European Heritage | 40 | 42 | 4 | 4 | 90

OUTCOME MEASURES:

1. Primary Outcome: Average Percentage Goal Volume Delivered Prior to Development of Intolerance for ITT Population
Description: The average percentage goal volume received via EN was defined as the percent of goal volume received via EN from the first study dose up to permanent discontinuation of EN. It is calculated as 100 multiplied by total volume received via EN during the on treatment period prior to intolerance divided by total prescribed volume. 'Prior to intolerance' means 'prior to start of intolerance treatment. One participant was missing for prior to start of intolerance treatment. The average percentage goal volume received via EN was assessed and comparison between Camicinal 50mg and placebo arm was performed. Adjusted mean and its 95% confidence interval (CI) were estimated and Analysis of Covariance (ANCOVA) model was used for analysis.
Time Frame: Up to Day 7
Population: Intension To Treat [ITT (exposed)] Population. ITT (exposed) Population comprised of all randomized participants who received at least of one dose of study treatment.
Measure: Mean (95% Confidence Interval); unit: Percentage of goal volume
Groups:
- Camicinal 50 mg: EN tolerant participants at Baseline were randomized to receive up to 7 doses of Camicinal (GSK962040) 50 mg once daily via NG tube.
- Placebo: EN tolerant participants at Baseline were randomized to receive up to 7 doses of Placebo drug once daily via NG tube.
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
Percentage of goal volume | 76.6 [67.0 to 86.3] | 67.7 [57.6 to 77.8]
Statistical Analysis 1: Comparison: Camicinal 50 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 8.9, 95% CI 2-sided [-5.1 to 22.9], Standard Error of Mean 7.02

2. Primary Outcome: Average Percentage Goal Volume Delivered Prior to Development of Intolerance for PP Population
Description: The average percentage goal volume received via EN was defined as the percent of goal volume received via EN from the first study dose up to permanent discontinuation of EN. It is calculated as 100 multiplied by total volume received via EN during the on treatment period prior to intolerance divided by total prescribed volume. 'Prior to intolerance' means 'prior to start of intolerance treatment. One participant was missing for prior to start of intolerance treatment. The average percentage goal volume received via EN was assessed and comparison between Camicinal 50mg and placebo arm was performed. Adjusted mean and its 95% CI were estimated and ANCOVA model was used for analysis.
Time Frame: Up to Day 7
Population: Per Protocol (PP) Population. PP Population comprised of all randomized participants who receive at least two doses of study treatment and have at least two days of evaluable nutritional data and also comply with the protocol.
Measure: Mean (95% Confidence Interval); unit: Percentage of goal volume
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 34 | 32
Percentage of goal volume | 76.6 [70.6 to 82.7] | 74.4 [68.2 to 80.6]
Statistical Analysis 1: Comparison: Camicinal 50 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-6.5 to 10.9], Standard Error of Mean 4.35

3. Secondary Outcome: Average Percentage Goal Calories Delivered Prior to Development of Intolerance
Description: The average percentage goal calories received via EN was defined as the percent of goal calories received via EN from the first study dose up to permanent discontinuation of EN. It is calculated as 100 multiplied by total calories received via EN during the on treatment period prior to intolerance divided by total prescribed calories. 'Prior to intolerance' means 'prior to start of intolerance treatment. The average percentage goal calories received via EN was assessed and comparison between Camicinal 50mg and placebo arm was performed. Adjusted mean and its 95% CI were estimated and ANCOVA model was used for analysis.
Time Frame: Up to Day 7
Population: ITT (exposed) Population
Measure: Mean (95% Confidence Interval); unit: Percentage of goal calories
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
Percentage of goal calories | 76.7 [67.0 to 86.3] | 67.8 [57.6 to 77.9]
Statistical Analysis 1: Comparison: Camicinal 50 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 8.9, 95% CI 2-sided [-5.1 to 22.9], Standard Error of Mean 7.03

4. Secondary Outcome: Average Percentage Goal Protein Delivered Prior to Development of Intolerance
Description: The average percentage goal protein received via EN was defined as the percent of goal protein received via EN from the first study dose up to permanent discontinuation of EN. It is calculated as 100 multiplied by total protein received via EN during the on treatment period prior to intolerance divided by total prescribed protein. 'Prior to intolerance' means 'prior to start of intolerance treatment. One participant was missing for prior to start of intolerance treatment. The average percentage goal protein received via EN was assessed and comparison between Camicinal 50mg and placebo arm was performed. Adjusted mean and its 95% CI were estimated and ANCOVA model was used for analysis.
Time Frame: Up to Day 7
Population: ITT (exposed) Population
Measure: Mean (95% Confidence Interval); unit: Percentage of goal protein
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
Percentage of goal protein | 76.3 [67.0 to 85.5] | 69.8 [60.0 to 79.5]
Statistical Analysis 1: Comparison: Camicinal 50 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 6.5, 95% CI 2-sided [-6.9 to 19.9], Standard Error of Mean 6.74

5. Secondary Outcome: Time to Delivery of 80 Percent Prescribed Calories Prior to Intolerance
Description: Time required for the delivery of 80 percent prescribed calories prior to intolerance was calculated using Kaplan-Meier estimates for time variable. Prior to intolerance was defined as prior to start of intolerance treatment. Participants who did not reach delivery of 80 percent prescribed calories were censored at the last day on which they received randomized treatment and with available nutritional data.
Time Frame: Up to Day 7
Population: ITT (exposed) Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
Days | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 3.0]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinaemia were categorized as SAE.
Time Frame: up to 23 days
Population: Safety Population. Safety Population comprised of all participants who received at least one dose one study treatment.
Measure: Number; unit: Participants
Groups:
- Baseline EN Tolerant: Placebo: Participants who were tolerant to EN feeding at Baseline received up to 7 doses of placebo drug once daily via NG tube. Participants who developed intolerance did not switch the treatment.
- Baseline EN Tolerant: Camicinal 50 mg: Participants who were tolerant to EN feeding at Baseline received up to 7 doses of Camicinal (GSK962040) 50 mg once daily via NG tube. participants who developed intolerance did not switch the treatment.
- Baseline EN Tolerant: Placebo/Camicinal 50 mg: Participants who were tolerant to EN feeding at Baseline received up to 7 doses of placebo drug once daily via NG tube. Participants who developed intolerance to EN feeding at any point up to dose 5 were switched to receive Camicinal 50 mg once daily.
- Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg: Participants who were tolerant to EN feeding at Baseline received up to 7 doses of either Camicinal (GSK962040) 50 mg once daily via NG tube. Participants who developed intolerance to EN feeding at any point up to dose 5 were switched to receive Metoclopramide 10 mg every 6 hrs via IV route.
- Baseline EN Intolerant: Camicinal 50 mg: Participant who were intolerant to EN feeding at Baseline received Camicinal (GSK962040) 50 mg once daily via NG tube.
- Baseline EN Intolerant: Metoclopramide 10 mg: Participant who were intolerant to EN feeding at Baseline received metoclopramide 10 mg every 6 Hrs. via IV route.
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
Participants
  AE | 9 | 13 | 2 | 2 | 0 | 3
  SAE | 1 | 4 | 0 | 0 | 0 | 2

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured at Baseline, Day 1, up to 6 hrs pre-dose on Day 2-7 and at follow-up (till 23 days). The Baseline value was considered to be the participant's last available assessment prior to randomized treatment. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, SBP and DBP were measured at Day 1 to Day 7 post-intolerance. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the standard deviation (SD) was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
millimeter of mercury (mmHg)
  DBP Day1; n= 23,33,1,3,0,0 | -1.1 (10.51) | -1.0 (9.84) | 5.0 (NA) — NA indicates that data were not available. | -2.0 (13.89) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  DBP Day2; n= 33,38,2,2,0,0 | 2.7 (12.77) | -0.2 (11.66) | -1.5 (NA) — NA indicates that data were not available. | 6.5 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  DBP Day3; n= 29,31,1,1,0,0 | 2.2 (12.12) | 1.7 (10.44) | 5.0 (NA) — NA indicates that data were not available. | -16.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  DBP Day4; n=25,27,0,0,0,0 | 2.9 (15.03) | 3.2 (13.37) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  DBP Day5; n= 22,23,0,0,0,0 | 5.3 (16.12) | -0.7 (15.66) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  DBP Day6; n= 18,19,0,0,0,0 | 2.6 (17.03) | 2.3 (15.86) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  DBP Day7; n= 14,14,0,0,0,0 | -4.6 (15.33) | -2.4 (13.89) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  DBP Intolerance Day1; n=1,0,3,3,3,3 | 7.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 9.3 (4.04) | -0.3 (11.27) | 11.0 (7.81) | 0.0 (14.42)
  DBP Intolerance Day2; n=0,0,2,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.5 (NA) — NA indicates that data were not available. | -12.0 (6.24) | 23.5 (17.71) | -4.0 (15.08)
  DBP Intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 10.5 (NA) — NA indicates that data were not available. | 6.3 (9.07) | 4.3 (8.39) | -0.5 (4.36)
  DBP Intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 9.0 (NA) — NA indicates that data were not available. | 15.5 (NA) — NA indicates that data were not available. | 11.7 (8.50) | -1.7 (9.24)
  DBP Intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -5.0 (NA) — NA indicates that data were not available. | 2.0 (NA) — NA indicates that data were not available. | 5.3 (4.51) | 1.7 (18.50)
  DBP Intolerance Day6; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 14.5 (NA) — NA indicates that data were not available. | -3.0 (NA) — NA indicates that data were not available. | 7.3 (4.62) | 13.7 (25.97)
  DBP Intolerance Day7; n= 0,0,0,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.7 (7.51) | 8.5 (NA) — NA indicates that data were not available.
  DBP Follow up; n= 27,28,3,3,4,2 | 9.1 (20.14) | 6.7 (13.70) | 23.0 (6.08) | 18.0 (4.58) | 4.0 (6.98) | 29.0 (NA) — NA indicates that data were not available.
  SBP Day1; n= 23,33,1,3,0,0 | -4.6 (19.58) | 1.0 (24.37) | 1.0 (NA) — NA indicates that data were not available. | 3.0 (23.64) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  SBP Day2; n= 33,38,2,2,0,0 | 3.7 (22.66) | 1.4 (23.55) | 12.5 (NA) — NA indicates that data were not available. | 16.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  SBP Day3; n= 29,31,1,1,0,0 | 5.1 (28.06) | 4.9 (25.00) | 6.0 (NA) — NA indicates that data were not available. | -16.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  SBP Day4; n= 25,27,0,0,0,0 | 7.6 (21.76) | 6.0 (30.02) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  SBP Day5; n= 22,23,0,0,0,0 | 11.3 (27.16) | -0.6 (34.31) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  SBP Day6; n= 18,19,0,0,0,0 | -1.6 (34.29) | -4.2 (33.26) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  SBP Day7; n= 14,14,0,0,0,0 | -2.5 (37.96) | -5.4 (24.47) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  SBP Intolerance Day1; n= 1,0,3,3,3,3 | -2.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 16.3 (12.66) | 1.7 (11.50) | 1.0 (13.08) | -4.7 (9.07)
  SBP Intolerance Day2; n= 0,0,2,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.5 (NA) — NA indicates that data were not available. | -9.3 (10.60) | 32.8 (31.06) | -4.0 (7.79)
  SBP Intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 11.0 (NA) — NA indicates that data were not available. | 16.3 (22.37) | 30.7 (12.22) | 13.0 (21.18)
  SBP Intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 19.5 (NA) — NA indicates that data were not available. | 22.0 (NA) — NA indicates that data were not available. | 43.0 (16.52) | -9.0 (12.29)
  SBP Intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 17.0 (NA) — NA indicates that data were not available. | 15.0 (NA) — NA indicates that data were not available. | 19.7 (24.79) | 8.7 (7.02)
  SBP Intolerance Day6; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 46.5 (NA) — NA indicates that data were not available. | 5.0 (NA) — NA indicates that data were not available. | 20.3 (21.73) | 10.7 (10.41)
  SBP Intolerance Day7; n= 0,0,0,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 22.0 (11.36) | 13.0 (NA) — NA indicates that data were not available.
  SBP follow up; n= 27,28,3,3,4,2 | -0.6 (25.75) | -1.4 (30.61) | 26.0 (17.58) | 3.0 (28.51) | 11.8 (18.14) | 14.0 (NA) — NA indicates that data were not available.

8. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: HR was measured at Baseline, Day 1, up to 6 hrs pre-dose on Day 2-7 and at follow-up (till Day 23). The Baseline value was considered to be the participant's last available assessment prior to randomized treatment. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, HR was measured at Day 1 to Day 7 post-intolerance. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
beats per minute (bpm)
  HR Day1; n= 23,33,1,3,0,0 | -4.0 (10.05) | 4.3 (14.13) | -5.0 (NA) — NA indicates that data were not available. | -0.7 (11.50) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  HR Day2; n= 34,38,2,2,0,0 | -1.6 (15.23) | -0.5 (14.61) | 4.5 (NA) — NA indicates that data were not available. | 5.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  HR Day3; n= 29,31, 1,1,0,0 | -0.0 (19.68) | 1.6 (12.93) | 26.0 (NA) — NA indicates that data were not available. | -21.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  HR Day4; n= 25,27,0,0,0,0 | -4.4 (19.84) | 2.1 (14.96) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  HR Day5; n= 22,23,0,0,0,0 | -3.0 (19.21) | 0.2 (17.17) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  HR Day6; n= 18,19,0,0,0,0 | -1.2 (22.26) | 1.4 (19.46) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  HR Day7; n= 14,14,,0,0,0,0 | -1.9 (19.17) | 0.6 (22.85) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  HR intolerance Day1; n= 1,0,3,3,3,3 | 6.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 19.7 (8.08) | -2.0 (13.89) | 1.3 (13.61) | 2.3 (2.52)
  HR intolerance Day2; n= 0,0,2,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 22.5 (NA) — NA indicates that data were not available. | -12.7 (16.62) | 9.0 (17.47) | 7.5 (11.90)
  HR intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 8.5 (NA) — NA indicates that data were not available. | 0.7 (12.50) | 6.3 (11.93) | 13.5 (12.48)
  HR intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 15.5 (NA) — NA indicates that data were not available. | -2.0 (NA) — NA indicates that data were not available. | 14.0 (19.47) | 5.3 (3.21)
  HR intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 9.0 (NA) — NA indicates that data were not available. | -3.0 (NA) — NA indicates that data were not available. | 19.0 (29.87) | 17.3 (16.17)
  HR intolerance Day6; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.5 (NA) — NA indicates that data were not available. | -1.0 (NA) — NA indicates that data were not available. | 19.7 (22.85) | 17.0 (11.53)
  HR intolerance Day7; n= 0,0,0,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 16.3 (20.50) | 16.0 (NA) — NA indicates that data were not available.
  HR follow up; n= 27,28,3,3,4,2 | 0.8 (19.76) | 2.7 (25.05) | 11.0 (15.87) | -2.0 (19.08) | 16.8 (21.73) | 27.0 (NA) — NA indicates that data were not available.

9. Secondary Outcome: Number of Participants With Maximum Increase From Baseline in Electrocardiogram (ECG) Values
Description: 12-lead ECGs was done at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7 and at follow up (till Day 23) that automatically calculates corrected QT (QTc), QTcF (QT duration corrected for heart rate by Fridericia's formula) and QTcB (QT duration corrected for heart rate by Bazett's formula) intervals. Three ECGs approximately 5 min apart were collected prior to dose 1and single recordings were made at other time points. On Day 1ECGs were collected at pre-dose (up to 6 hrs) and 2 hr post treatment. Number of participants with maximum increase from Baseline were collected and participants showed increase in 3 parameters namely QTc, QTcB and QTcF. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles).
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
Participants
  Day 1; QTc <= 60; n= 10,5,0,1,0,0 | 10 | 5 | 0 | 1 | 0 | 0
  Day 1; QTc >60; n= 10,5,0,1,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1; QTcB <=60; n= 23,28,3,2,0,0 | 23 | 27 | 3 | 2 | 0 | 0
  Day 1; QTcB >60; n= 23,28,3,2,0,0 | 0 | 1 | 0 | 0 | 0 | 0
  Day 1; QTcF <=60; n= 23,28,3,2,0,0 | 23 | 27 | 3 | 2 | 0 | 0
  Day 1; QTcF >60; n= 23,28,3,2,0,0 | 0 | 1 | 0 | 0 | 0 | 0
  Day 2; QTc <= 60; n= 8,7,0,1,0,0 | 8 | 7 | 0 | 1 | 0 | 0
  Day 2; QTc >60; n= 8,7,0,1,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 2; QTcB <=60; n= 23,28,2,1,0,0 | 23 | 26 | 2 | 1 | 0 | 0
  Day 2; QTcB >60; n= 23,28,2,1,0,0 | 0 | 2 | 0 | 0 | 0 | 0
  Day 2; QTcF <=60; n= 23,28,2,1,0,0 | 23 | 27 | 2 | 1 | 0 | 0
  Day 2; QTcF >60; n= 23,28,2,1,0,0 | 0 | 1 | 0 | 0 | 0 | 0
  Day 3; QTc <= 60; n= 7,6,0,1,0,0 | 7 | 6 | 0 | 1 | 0 | 0
  Day 3; QTc >60; n= 7,6,0,1,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 3; QTcB <=60; n= 19,21,1,0,0 | 18 | 21 | 1 | 0 | 0 | 0
  Day 3; QTcB >60; n= 19,21,1,0,0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 3; QTcF; <=60; n= 19,21,1,0,0,0 | 19 | 21 | 1 | 0 | 0 | 0
  Day 3; QTcF; >60; n= 19,21,1,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4; QTc; <=60; n= 7,5,0,0,0,0 | 7 | 5 | 0 | 0 | 0 | 0
  Day 4; QTc; >60; n= 7,5,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4; QTcB; <=60; n= 16,19,0,0,0,0 | 16 | 19 | 0 | 0 | 0 | 0
  Day 4; QTcB; >60; n= 16,19,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4; QTcF; <=60; n= 16,19,0,0,0,0 | 16 | 19 | 0 | 0 | 0 | 0
  Day 4; QTcF; >60; n= 16,19,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5; QTc; <=60; n= 7,5,0,0,0,0 | 7 | 5 | 0 | 0 | 0 | 0
  Day 5; QTc; >60; n= 7,5,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5; QTcB; <=60; n= 14,17,0,0,0,0 | 14 | 17 | 0 | 0 | 0 | 0
  Day 5; QTcB; >60; n= 14,17,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5; QTcF; <=60; n= 14,17,0,0,0,0 | 14 | 16 | 0 | 0 | 0 | 0
  Day 5; QTcF; >60; n= 14,17,0,0,0,0 | 0 | 1 | 0 | 0 | 0 | 0
  Day 6; QTc; <=60; n= 5,5,0,0,0,0 | 5 | 5 | 0 | 0 | 0 | 0
  Day 6; QTc; >60; n= 5,5,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 6; QTcB; <=60; n= 11,14,0,0,0,0 | 11 | 14 | 0 | 0 | 0 | 0
  Day 6; QTcB; >60; n= 11,14,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 6; QTcF; <=60; n= 11,14,0,0,0,0 | 11 | 14 | 0 | 0 | 0 | 0
  Day 6; QTcF; >60; n= 11,14,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7; QTc; <=60; n= 5,4,0,0,0,0 | 5 | 4 | 0 | 0 | 0 | 0
  Day 7; QTc; >60; n= 5,4,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7; QTcB; <=60; n= 8,11,0,0,0,0 | 8 | 11 | 0 | 0 | 0 | 0
  Day 7; QTcB; >60; n= 8,11,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7; QTcF; <=60; n= 8,11,0,0,0,0 | 8 | 11 | 0 | 0 | 0 | 0
  Day 7; QTcF; >60; n= 8,11,0,0,0,0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow up; QTc; <=60; n= 6,4,0,1,1,1 | 6 | 4 | 0 | 1 | 1 | 1
  Follow up; QTc; >60; n= 6,4,0,1,1,1 | 0 | 0 | 0 | 0 | 0 | 0
  Follow up; QTcB; <=60; n= 10,13,2,2,3,1 | 9 | 13 | 2 | 2 | 3 | 1
  Follow up; QTcB; >60; n= 10,13,2,2,3,1 | 1 | 0 | 0 | 0 | 0 | 0
  Follow up; QTcF;<=60; n= 10,13,2,2,2,1 | 9 | 13 | 2 | 2 | 2 | 1
  Follow up; QTcF; >60; n= 10,13,2,2,2,1 | 1 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 1; QTc; <=60; n=0,0,0,1,1,2 | 0 | 0 | 0 | 1 | 1 | 2
  Intolerance Day 1; QTc; >60; n= 0,0,0,1,1,2 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 1; QTcB; <=60; n= 0,0,3,2,3,1 | 0 | 0 | 3 | 2 | 3 | 1
  Intolerance Day 1; QTcB; >60; n= 0,0,3,2,3,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 1; QTcF; <=60; n= 0,0,3,2,3,1 | 0 | 0 | 3 | 2 | 3 | 1
  Intolerance Day 1; QTcF; >60; n= 0,0,3,2,3,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 2; QTc; <=60; n= 0,0,0,1,1,2 | 0 | 0 | 0 | 1 | 1 | 2
  Intolerance Day 2; QTc; >60; n= 0,0,0,1,1,2 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 2; QTcB; <=60; n= 0,0,3,2,2,1 | 0 | 0 | 3 | 2 | 2 | 1
  Intolerance Day 2; QTcB; >60; n= 0,0,3,2,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 2; QTcF; <=60; n= 0,0,3,2,2,1 | 0 | 0 | 3 | 2 | 2 | 1
  Intolerance Day 2; QTcF; >60; n= 0,0,3,2,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 3; QTc; <=60; n= 0,0,0,1,1,3 | 0 | 0 | 0 | 1 | 1 | 3
  Intolerance Day 3; QTc; >60; n= 0,0,0,1,1,3 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 3; QTcB; <=60; n= 0,0,2,2,2,1 | 0 | 0 | 2 | 2 | 2 | 1
  Intolerance Day 3; QTcB; >60; n= 0,0,2,2,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 3; QTcF; <=60; n= 0,0,2,2,2,1 | 0 | 0 | 2 | 2 | 2 | 1
  Intolerance Day 3; QTcF; >60; n= 0,0,2,2,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 4; QTc; <=60; n= 0,0,0,1,1,2 | 0 | 0 | 0 | 1 | 1 | 2
  Intolerance Day 4; QTc; >60; n= 0,0,0,1,1,2 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 4; QTcB; <=60; n= 0,0,2,1,2,1 | 0 | 0 | 2 | 1 | 2 | 1
  Intolerance Day 4; QTcB; >60; n= 0,0,2,1,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 4; QTcF; <=60; n= 0,0,2,1,2,1 | 0 | 0 | 2 | 1 | 2 | 1
  Intolerance Day 4; QTcF; >60; n= 0,0,2,1,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 5; QTc; <=60; n=0,0,0,0,1,2 | 0 | 0 | 0 | 0 | 1 | 1
  Intolerance Day 5; QTc; >60; n= 0,0,0,0,1,2 | 0 | 0 | 0 | 0 | 0 | 1
  Intolerance Day 5; QTcB; <=60; n= 0,0,1,1,2,1 | 0 | 0 | 1 | 1 | 2 | 1
  Intolerance Day 5; QTcB; >60; n= 0,0,1,1,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 5; QTcF; <=60; n= 0,0,1,1,2,1 | 0 | 0 | 1 | 1 | 2 | 1
  Intolerance Day 5; QTcF; >60; n= 0,0,1,1,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 6; QTc; <=60; n= 0,0,0,0,1,2 | 0 | 0 | 0 | 0 | 1 | 2
  Intolerance Day 6; QTc; >60; n= 0,0,0,0,1,2 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 6; QTcB; <=60; n= 0,0,2,1,2,1 | 0 | 0 | 2 | 1 | 2 | 1
  Intolerance Day 6; QTcB; >60; n= 0,0,2,1,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 6; QTcF; <=60; n= 0,0,2,1,2,1 | 0 | 0 | 2 | 1 | 2 | 1
  Intolerance Day 6; QTcF; >60; n= 0,0,2,1,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 7; QTc; <=60; n= 0,0,0,0,1,1 | 0 | 0 | 0 | 0 | 1 | 1
  Intolerance Day 7; QTc; >60; n= 0,0,0,0,1,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 7; QTcB; <=60; n= 0,0,0,0,2,1 | 0 | 0 | 0 | 0 | 2 | 1
  Intolerance Day 7; QTcB; >60; n= 0,0,0,0,2,1 | 0 | 0 | 0 | 0 | 0 | 0
  Intolerance Day 7; QTcF; <=60; n= 0,0,0,0,2,1 | 0 | 0 | 0 | 0 | 2 | 1
  Intolerance Day 7; QTcF; >60; n= 0,0,0,0,2,1 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Albumin and Total Protein Levels
Description: Blood samples were collected to evaluate change from Baseline in albumin and total protein values at Baseline, Day 2-7 and follow-up (till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
Gram per liter (g/L)
  Albumin Day 2; n=1,1,0,0,0,0 | 4.00 (NA) — NA indicates that data were not available. | -1.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin; Day 3; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -3.50 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin Day 4; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -3.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin Day 5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.50 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin Day 6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -4.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin Day 7; n= 13,11,0,0,0,0 | 0.98 (6.202) | 0.64 (6.795) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin intolerance Day 2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.00 (NA) — NA indicates that data were not available.
  Albumin intolerance Day 3; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -3.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin intolerance Day 4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin intolerance Day 6; n= 0,0,1,1,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.00 (NA) — NA indicates that data were not available. | -3.00 (NA) — NA indicates that data were not available. | 11.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Albumin intolerance Day 7; n= 0,0,1,0,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -6.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.00 (NA) — NA indicates that data were not available. | 1.20 (NA) — NA indicates that data were not available.
  Albumin follow up; n= 18,17,3,3,4,2 | 5.81 (5.827) | 4.59 (6.526) | 4.73 (5.139) | 8.33 (3.512) | 5.25 (4.500) | 2.30 (NA) — NA indicates that data were not available.
  Total protein Day 2; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -3.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total protein Day 3; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 9.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total protein Day 5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 7.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total protein Day 6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -2.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total protein Day 7; n= 10,11,0,0,0,0 | 10.06 (9.663) | 3.21 (4.733) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total protein intolerance Day 2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.00 (NA) — NA indicates that data were not available.
  Total protein intolerance Day 3; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 6.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total protein intolerance Day 4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 14.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total protein intolerance Day 6; n= 0,0,1,1,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 22.00 (NA) — NA indicates that data were not available. | 8.00 (NA) — NA indicates that data were not available. | 2.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total protein intolerance Day 7; n= 0,0,1,0,1,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 2.00 (NA) — NA indicates that data were not available. | 10.75 (NA) — NA indicates that data were not available.
  Total protein follow up; n= 15,16,3,3,4,2 | 16.27 (13.598) | 16.43 (10.423) | 20.77 (2.250) | 22.33 (7.234) | 4.50 (17.540) | 18.60 (NA) — NA indicates that data were not available.

11. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (Alk. Phosph.), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Gamma Glutamyl Transferase (GGT) Levels
Description: Blood samples were collected to evaluate change from Baseline in alk.phosp., ALT, AST and GGT values at Baseline, Day 1- Day 7 and follow up (till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International Unit per liter (IU/L)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
International Unit per liter (IU/L)
  Alk. phosp. Day 2; n= 32,34,2,2,0,0 | 2.7 (19.60) | 7.9 (19.39) | 2.5 (NA) — NA indicates that data were not available. | -2.5 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  ALk. phosp. Day 3; n= 28,28,1,1,0,0 | -1.5 (42.47) | 21.5 (27.98) | 43.0 (NA) — NA indicates that data were not available. | 19.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Alk. phosp. Day 4; n= 25,25,0,0,0,0 | 11.2 (24.62) | 25.4 (38.55) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Alk. phsp Day5; n= 22,23,0,0,0,0 | 14.2 (33.14) | 36.6 (49.26) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Alk. phsp Day6; n= 18,19,0,0,0,0 | 13.4 (36.49) | 53.6 (78.10) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Alk. phsp. Day7; n= 14,13,0,0,0,0 | 13.9 (33.93) | 74.6 (93.12) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Alk. phosp. intolerance Day1; n= 1,0,2,3,0,0 | 24.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 38.0 (NA) — NA indicates that data were not available. | 11.7 (14.19) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Alk. phosp. intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 37.7 (37.55) | 20.0 (10.44) | 5.8 (13.10) | 18.0 (35.13)
  Alk. phosp. intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 22.0 (NA) — NA indicates that data were not available. | 23.0 (17.69) | -5.0 (21.07) | 39.3 (38.34)
  Alk. phosp. intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 47.0 (NA) — NA indicates that data were not available. | 56.5 (NA) — NA indicates that data were not available. | 2.3 (23.07) | 56.0 (45.13)
  Alk. phosp. intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 46.5 (NA) — NA indicates that data were not available. | 67.0 (NA) — NA indicates that data were not available. | 35.5 (NA) — NA indicates that data were not available. | 81.3 (16.56)
  Alk. phosp. intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 51.5 (NA) — NA indicates that data were not available. | 56.0 (NA) — NA indicates that data were not available. | 29.7 (46.82) | 53.5 (NA) — NA indicates that data were not available.
  Alk. phosp. intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 76.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 25.0 (47.16) | 65.5 (NA) — NA indicates that data were not available.
  Alk.phosp. follow up; n= 17,20,3,2,4,2 | 32.4 (85.80) | 76.0 (147.05) | 274.0 (272.24) | 71.5 (NA) — NA indicates that data were not available. | 77.5 (86.03) | 110.5 (NA) — NA indicates that data were not available.
  ALT Day 2; n= 32,35,2,2,0,0 | -1.9 (16.07) | 2.0 (16.53) | -19.5 (NA) — NA indicates that data were not available. | -1.5 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  ALT Day 3; n= 29,30,1,1,0,0 | -2.8 (37.00) | 7.2 (27.49) | 6.0 (NA) — NA indicates that data were not available. | 8.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  ALT Day 4; n= 25,25,0,0,0,0 | -4.0 (53.27) | 7.0 (29.81) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  ALT Day 5; n= 22,23,0,0,0,0 | 0.4 (70.15) | 6.7 (34.80) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  ALT Day 6; n= 18,19,0,0,0,0 | 0.1 (84.99) | 8.5 (44.37) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  ALT Day 7; n= 14,13,0,0,0,0 | -5.4 (95.92) | 14.8 (75.08) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  ALT intolerance Day 1; n= 1,0,2,3,0,0 | 1.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -2.0 (NA) — NA indicates that data were not available. | 9.3 (15.50) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  ALT intolerance Day 2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -25.3 (38.37) | 14.0 (7.55) | 6.5 (9.47) | 28.3 (61.24)
  ALT intolerance Day 3; n= n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -68.0 (NA) — NA indicates that data were not available. | 14.3 (9.61) | 8.3 (10.50) | 34.5 (55.70)
  ALT intolerance Day 4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -77.0 (NA) — NA indicates that data were not available. | 41.5 (NA) — NA indicates that data were not available. | 24.3 (30.09) | 118.3 (65.55)
  ALT intolerance Day 5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -81.0 (NA) — NA indicates that data were not available. | 50.0 (NA) — NA indicates that data were not available. | 34.0 (47.66) | 193.7 (59.58)
  ALT intolerance Day 6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -75.5 (NA) — NA indicates that data were not available. | 45.0 (NA) — NA indicates that data were not available. | 44.3 (57.87) | 189.0 (NA) — NA indicates that data were not available.
  ALT intolerance Day 7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -20.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 35.3 (49.17) | 136.5 (NA) — NA indicates that data were not available.
  ALT follow up; n= n= 18,20,3,3,4,2 | -4.6 (93.05) | 29.2 (62.61) | -59.7 (68.73) | 50.7 (62.74) | 58.8 (56.20) | 29.5 (NA) — NA indicates that data were not available.
  AST Day 2; n= 31,34,2,1,0,0 | -8.742 (40.5873) | 0.118 (23.3936) | -36.500 (NA) — NA indicates that data were not available. | -9.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  AST Day3; n= 28,29,1,1,0,0 | -11.500 (65.8598) | -4.828 (39.6260) | -18.000 (NA) — NA indicates that data were not available. | 16.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  AST Day4; n= 23,23,0,0,0,0 | -14.348 (83.2317) | -14.870 (60.7329) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  AST Day5; n= 22,22,0,0,0,0 | -11.518 (88.6693) | -14.318 (66.3672) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  AST Day6; n= 18,18,0,0,0,0 | -18.222 (99.4494) | -10.944 (75.4262) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  AST Day7; n= 13,12,0,0,0,0 | -29.538 (115.0454) | -11.417 (104.7147) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  AST intolerance Day1; n= 1,0,2,1,0,0 | -11.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -50.000 (NA) — NA indicates that data were not available. | 1.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  AST intolerance Day2; n= 0,0,3,1,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -69.000 (19.0000) | 28.000 (NA) — NA indicates that data were not available. | 8.500 (15.1548) | 6.000 (8.0829)
  AST intolerance Day3; n= 0,0,2,2,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -96.000 (NA) — NA indicates that data were not available. | 22.000 (NA) — NA indicates that data were not available. | 0.333 (2.0817) | 20.250 (16.8795)
  AST intolerance Day4; n= 0,0,1,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -66.000 (NA) — NA indicates that data were not available. | 49.500 (NA) — NA indicates that data were not available. | 22.000 (32.1870) | 126.333 (91.1939)
  AST intolerance Day5; n= 0,0,1,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -63.000 (NA) — NA indicates that data were not available. | 46.000 (NA) — NA indicates that data were not available. | 19.000 (27.0555) | 281.000 (NA) — NA indicates that data were not available.
  AST intolerance Day6; n= 0,0,1,1,3,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -46.000 (NA) — NA indicates that data were not available. | 30.000 (NA) — NA indicates that data were not available. | 18.667 (17.4738) | 374.000 (NA) — NA indicates that data were not available.
  AST intolerance Day7; n= 0,0,1,0,3,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -64.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.333 (10.0167) | 171.000 (NA) — NA indicates that data were not available.
  AST follow up; n= 17,20,3,2,4,2 | -33.412 (99.3511) | 4.500 (82.3551) | -110.333 (24.7049) | 8.500 (NA) — NA indicates that data were not available. | 47.000 (81.5475) | -3.500 (NA) — NA indicates that data were not available.
  GGT Day2; n= 32,34,2,2,0,0 | 7.4 (38.77) | 19.3 (41.39) | 5.5 (NA) — NA indicates that data were not available. | 8.5 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  GGT Day3; n= 28,28,1,1,0,0 | 13.4 (95.74) | 49.8 (62.30) | 75.0 (NA) — NA indicates that data were not available. | 74.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  GGT Day4; n= 24,24,0,0,0,0 | 54.8 (77.91) | 51.0 (52.82) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  GGT Day5; n= 22,22,0,0,0,0 | 81.7 (106.54) | 82.1 (83.82) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  GGT Day6; n= 18,18,0,0,0,0 | 100.1 (150.79) | 100.3 (104.52) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  GGT Day7; n= 14,12,0,0,0,0 | 85.6 (99.69) | 156.0 (156.59) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  GGT intolerance Day1; n= 1,0,2,3,0,0 | 43.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 66.0 (NA) — NA indicates that data were not available. | 41.7 (52.37) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  GGT intolerance Day2; n= 0,0,3,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 51.0 (34.18) | 59.0 (47.57) | 21.0 (11.79) | 25.3 (41.42)
  GGT intolerance Day3; n= 0,0,2,3,2,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 46.5 (NA) — NA indicates that data were not available. | 89.0 (73.08) | 28.5 (NA) — NA indicates that data were not available. | 65.5 (86.38)
  GGT intolerance Day4; n= 0,0,2,2,2,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 153.0 (NA) — NA indicates that data were not available. | 216.0 (NA) — NA indicates that data were not available. | 45.5 (NA) — NA indicates that data were not available. | 196.7 (129.53)
  GGT intolerance Day5; n= 0,0,2,1,2,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 201.5 (NA) — NA indicates that data were not available. | 223.0 (NA) — NA indicates that data were not available. | 82.5 (NA) — NA indicates that data were not available. | 269.3 (60.07)
  GGT intolerance Day6; n= 0,0,2,1,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 249.5 (NA) — NA indicates that data were not available. | 218.0 (NA) — NA indicates that data were not available. | 116.5 (NA) — NA indicates that data were not available. | 399.5 (NA) — NA indicates that data were not available.
  GGT intolerance Day7; n= 0,0,1,0,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 400.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 118.5 (NA) — NA indicates that data were not available. | 590.0 (NA) — NA indicates that data were not available.
  GGT follow up; n= 18,20,3,3,3,2 | 84.6 (158.30) | 84.9 (164.37) | 140.0 (89.87) | 78.0 (29.87) | 224.0 (24.56) | 216.0 (NA) — NA indicates that data were not available.

12. Secondary Outcome: Change From Baseline in Total and Direct Bilirubin, Creatinine and Uric Acid Levels
Description: Blood samples were collected to evaluate change from Baseline in total and direct bilirubin, creatinine and uric acid values at Baseline, Day 2- Day 7 and at follow up (Till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: micromoles per Liter (µmol/L)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
micromoles per Liter (µmol/L)
  Direct bilirubin; Day 2; n= 28,26,2,1,0,0 | -1.246 (3.7551) | 0.088 (2.8035) | 0.800 (NA) — NA indicates that data were not available. | 1.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Direct bilirubin Day3; n= 25,23,1,1,0,0 | -1.512 (3.8420) | -0.126 (3.2325) | 25.300 (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Direct bilirubin; Day4; n= 19,18,0,0,0,0 | 0.700 (6.2765) | 0.172 (1.3323) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Direct bilirubin; Day5; n= 17,15,0,0,0,0 | 1.482 (10.6636) | -1.007 (4.7148) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Direct bilirubin; Day6; n= 13,12,0,0,0,0 | 1.031 (9.5551) | -0.583 (2.5933) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Direct bilirubin; Day7; n= 10,7,0,0,0,0 | 3.240 (16.6513) | -1.214 (4.9229) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Direct bilirubin; intolerance Day1; n= 1,0,2,2,0,0 | 0.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.100 (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Direct bilirubin; intolerance Day2; n= 0,0,2,1,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.100 (NA) — NA indicates that data were not available. | 1.000 (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | 1.700 (NA) — NA indicates that data were not available.
  Direct bilirubin; intolerance Day3; n= 0,0,1,2,1,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.000 (NA) — NA indicates that data were not available. | 0.500 (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | 12.167 (19.9144)
  Direct bilirubin; intolerance Day4; n= 0,0,1,1,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 5.000 (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | 0.500 (NA) — NA indicates that data were not available. | 4.800 (NA) — NA indicates that data were not available.
  Direct bilirubin; intolerance Day5; n= 0,0,1,1,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.000 (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | -1.050 (NA) — NA indicates that data were not available.
  Direct bilirubin; intolerance Day6; n=0,0,1,0,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.500 (NA) — NA indicates that data were not available. | -7.100 (NA) — NA indicates that data were not available.
  Direct bilirubin; intolerance Day7; n= 0,0,1,0,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.500 (NA) — NA indicates that data were not available. | -8.050 (NA) — NA indicates that data were not available.
  Direct bilirubin; follow up; n= 13,15,2,2,2,2 | -1.969 (3.6992) | -1.507 (4.2699) | 0.100 (NA) — NA indicates that data were not available. | -0.500 (NA) — NA indicates that data were not available. | 16.000 (NA) — NA indicates that data were not available. | -15.000 (NA) — NA indicates that data were not available.
  Total bilirubin; Day2; n= 32,35,2,2,0,0 | -1.172 (4.4060) | 0.326 (4.0836) | -1.350 (NA) — NA indicates that data were not available. | 0.500 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total bilirubin; Day3; n= 29,30,1,1,0,0 | -1.038 (3.6544) | -0.660 (7.4569) | 25.700 (NA) — NA indicates that data were not available. | 1.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total bilirubin; Day4; n= 25,25,0,0,0,0 | 0.496 (8.6799) | -0.840 (7.1559) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total bilirubin; Day5; n=22,22,0,0,0,0 | 1.168 (12.9402) | -1.055 (6.5842) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total bilirubin; Day6; n= 18,19,0,0,0,0 | 0.772 (11.3841) | -1.558 (7.2077) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total bilirubin; Day7; n= 14,12,0,0,0,0 | 2.964 (17.7740) | -3.133 (10.6133) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total bilirubin; intolerance Day1; n= 1,0,2,3,0,0 | -1.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 6.700 (NA) — NA indicates that data were not available. | 0.667 (2.5166) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Total bilirubin; intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.100 (4.5310) | 1.000 (2.6458) | -0.075 (1.0751) | 4.675 (6.6249)
  Total bilirubin; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 5.000 (NA) — NA indicates that data were not available. | 0.333 (3.2146) | 0.167 (0.7638) | 10.475 (19.6274)
  Total bilirubin; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 5.500 (NA) — NA indicates that data were not available. | 3.000 (NA) — NA indicates that data were not available. | 0.833 (2.7538) | 3.333 (4.9329)
  Total bilirubin; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.500 (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | 0.633 (2.0984) | -1.100 (4.2579)
  Total bilirubin; intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.500 (NA) — NA indicates that data were not available. | -1.000 (NA) — NA indicates that data were not available. | 0.000 (2.0000) | -8.050 (NA) — NA indicates that data were not available.
  Total bilirubin; intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.800 (2.3065) | -9.250 (NA) — NA indicates that data were not available.
  Total bilirubin; follow up; n= 19,20,3,2,4,2 | -1.263 (4.8442) | -1.805 (8.3199) | -0.467 (8.2978) | -2.000 (NA) — NA indicates that data were not available. | 10.850 (25.5152) | -17.000 (NA) — NA indicates that data were not available.
  Creatinine; Day2; n= 33,37,2,2,0,0 | -2.1818 (9.34898) | -1.4281 (28.09838) | -13.5000 (NA) — NA indicates that data were not available. | -5.0000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Creatinine; Day3; n= 29,31,1,1,0,0 | -4.2724 (16.74713) | -5.0323 (22.15774) | -3.0000 (NA) — NA indicates that data were not available. | -3.0000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Creatinine; Day4; n= 25,26,0,0,0,0 | -6.2400 (14.29534) | -3.6923 (32.58683) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Creatinine; Day5; n= 22,22,0,0,0,0 | -7.0909 (16.52389) | 1.5909 (52.62053) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Creatinine; Day6; n= 18,19,0,0,0,0 | -7.5000 (21.34658) | 19.7895 (83.59198) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Creatinine; Day7; n= 14,15,0,0,0,0 | -7.5714 (26.46831) | 6.4000 (78.29322) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Creatinine; intolerance Day1; n= 1,0,2,3,0,0 | -11.0000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.5000 (NA) — NA indicates that data were not available. | -1.6667 (3.51188) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Creatinine; intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.6667 (10.06645) | -5.6667 (5.13160) | 5.7500 (20.79062) | -1.5000 (11.90238)
  Creatinine; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -5.5000 (NA) — NA indicates that data were not available. | -4.6667 (5.50757) | 3.3333 (36.29509) | -21.5000 (22.60531)
  Creatinine; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.0000 (NA) — NA indicates that data were not available. | -6.0000 (NA) — NA indicates that data were not available. | -13.0000 (30.34798) | -14.0000 (22.60531)
  Creatinine; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -23.0000 (NA) — NA indicates that data were not available. | -10.0000 (NA) — NA indicates that data were not available. | -11.3333 (27.15388) | -16.6667 (20.59935)
  Creatinine; intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -28.5000 (NA) — NA indicates that data were not available. | -10.0000 (NA) — NA indicates that data were not available. | -12.3333 (34.93327) | -32.5000 (NA) — NA indicates that data were not available.
  Creatinine; intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -50.0000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -4.3333 (48.33563) | -34.0000 (NA) — NA indicates that data were not available.
  Creatinine; follow up; n= 25,28,3,3,4,2 | -5.8400 (20.46477) | 11.6786 (103.9060) | -34.0000 (13.52775) | -4.0000 (11.35782) | -12.0000 (24.17988) | -39.0000 (NA) — NA indicates that data were not available.
  Uric acid; Day3; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -70.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Uric acid; Day5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -20.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Uric acid; Day6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 282.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Uric acid; Day7; 11,11,0,0,0,0 | -20.18 (108.547) | -15.36 (152.550) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Uric acid; intolerance Day2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -3640.00 (NA) — NA indicates that data were not available.
  Uric acid; intolerance Day3; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -20.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Uric acid; intolerance Day4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 153.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Uric acid; intolerance Day6; n= 0,0,0,1,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -20.00 (NA) — NA indicates that data were not available. | 27.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Uric acid; intolerance Day7; n= 0,0,1,0,1,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -270.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -100.00 (NA) — NA indicates that data were not available. | 60.40 (NA) — NA indicates that data were not available.
  Uric acid follow up; n= 15,14,2,3,3,2 | 60.47 (96.092) | 58.36 (144.871) | -25.50 (NA) — NA indicates that data were not available. | 115.67 (106.228) | 72.33 (118.095) | 1076.90 (NA) — NA indicates that data were not available.

13. Secondary Outcome: Change From Baseline in Calcium, Chloride, Carbon Dioxide, Glucose, Potassium, Sodium, Blood Urea Nitrogen (BUN) Values
Description: Blood samples were collected to evaluate change from Baseline in calcium, chloride, carbon dioxide, glucose, potassium, sodium, BUN values at Baseline, up to Day 7 and follow up (till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: millimol per liter (mmol/L)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
millimol per liter (mmol/L)
  Calcium; Day 2; n= 1,2,0,0,0,0 | -0.0500 (NA) — NA indicates that data were not available. | 0.0000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; Day 3; n= 1,2,0,0,0,0 | 0.0200 (NA) — NA indicates that data were not available. | 0.1300 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; Day 4; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.0800 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; Day 5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.1500 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; Day 6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.0100 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; Day 7; n= 12,12,0,0,0,0 | 0.2208 (0.29222) | 0.0733 (0.12390) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; intolerance Day 2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.0400 (NA) — NA indicates that data were not available.
  Calcium; intolerance Day 3; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.3400 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; intolerance Day 4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.2100 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; intolerance Day 6; n= 0,0,1,1,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.3400 (NA) — NA indicates that data were not available. | 0.3600 (NA) — NA indicates that data were not available. | 0.4300 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Calcium; intolerance Day 7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.0700 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.2000 (0.36661) | 0.0200 (NA) — NA indicates that data were not available.
  Calcium; follow up; n= 19,18,3,3,4,2 | 0.2821 (0.19277) | 0.2483 (0.24957) | 0.2667 (0.02517) | 0.4767 (0.22008) | 0.2850 (0.39467) | 0.2050 (NA) — NA indicates that data were not available.
  Chloride; Day 2; n= 33,37,2,2,0,0 | -1.2 (2.66) | -0.6 (3.38) | -2.0 (NA) — NA indicates that data were not available. | -0.5 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Chloride; Day3; n= 28,31,1,1,0,0 | -1.5 (3.38) | -1.3 (4.26) | -5.0 (NA) — NA indicates that data were not available. | -7.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Chloride; Day4 ; n= 25,26,0,0,0,0 | -2.3 (3.93) | -1.8 (5.86) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Chloride; Day5; n= 22,23,0,0,0,0 | -3.4 (5.64) | -2.6 (6.93) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Chloride; Day 6; n= 18,19,0,0,0,0 | -4.1 (7.28) | -4.8 (7.52) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Chloride; Day7; n= 14,15,0,0,0,0 | -4.3 (7.49) | -3.1 (7.14) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Chloride intolerance Day 1; n= 1,0,2,3,0,0 | -1.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -6.0 (NA) — NA indicates that data were not available. | -3.7 (9.07) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Chloride intolerance Day 2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -5.3 (3.21) | -4.3 (8.50) | 0.5 (1.00) | -0.5 (3.42)
  Chloride intolerance Day 3; n= 0,0,2,3,2,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -6.5 (NA) — NA indicates that data were not available. | -6.0 (9.54) | 0.0 (NA) — NA indicates that data were not available. | -2.3 (4.99)
  Chloride intolerance Day 4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -5.0 (NA) — NA indicates that data were not available. | -11.0 (NA) — NA indicates that data were not available. | 2.3 (0.58) | -4.0 (7.00)
  Chloride intolerance Day 5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.5 (NA) — NA indicates that data were not available. | -2.0 (NA) — NA indicates that data were not available. | 4.3 (1.53) | -4.7 (4.51)
  Chloride intolerance Day 6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0 (NA) — NA indicates that data were not available. | -4.0 (NA) — NA indicates that data were not available. | 5.7 (2.08) | -4.0 (NA) — NA indicates that data were not available.
  Chloride intolerance Day 7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.3 (4.04) | -6.5 (NA) — NA indicates that data were not available.
  Chloride follow up; n= 22,23,3,3,3,2 | -6.1 (6.71) | -4.6 (6.27) | -7.3 (5.51) | -11.0 (5.57) | -7.0 (6.08) | -8.5 (NA) — NA indicates that data were not available.
  Carbon dioxide; Day 2; n= 32,36,2,2,0,0 | 3.31 (10.711) | 0.21 (3.770) | 2.50 (NA) — NA indicates that data were not available. | 1.50 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Carbon dioxide; Day 3; n= 27,31,1,1,0,0 | 1.64 (2.274) | 0.93 (6.406) | 6.00 (NA) — NA indicates that data were not available. | 3.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Carbon dioxide; Day 4; n= 24,25,0,0,0,0 | 0.43 (3.958) | 1.58 (8.054) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Carbon dioxide; Day 5; n= 20,22,0,0,0,0 | -0.16 (3.797) | 1.64 (7.631) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Carbon dioxide; Day 6; n= 16,16,0,0,0,0 | 0.64 (5.728) | 3.63 (5.308) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Carbon dioxide; Day 7; n= 12,13,0,0,0,0 | 0.98 (5.774) | 3.05 (4.945) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Carbon dioxide; intolerance Day1; n= 1,0,2,3,0,0 | 2.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.50 (NA) — NA indicates that data were not available. | 0.33 (2.082) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Carbon dioxide; intolerance Day2; n= 0,0,3,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.67 (1.528) | 0.33 (0.577) | -2.00 (3.000) | 0.93 (2.844)
  Carbon dioxide; intolerance Day3; n= 0,0,2,3,2,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 6.50 (NA) — NA indicates that data were not available. | 1.67 (2.309) | 1.00 (NA) — NA indicates that data were not available. | 2.80 (5.071)
  Carbon dioxide; intolerance Day4; n= 0,0,2,2,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 5.50 (NA) — NA indicates that data were not available. | 2.50 (NA) — NA indicates that data were not available. | 2.00 (NA) — NA indicates that data were not available. | 4.40 (NA) — NA indicates that data were not available.
  Carbon dioxide; intolerance Day5; n= 0,0,2,1,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 6.50 (NA) — NA indicates that data were not available. | 4.00 (NA) — NA indicates that data were not available. | 3.00 (NA) — NA indicates that data were not available. | 4.75 (NA) — NA indicates that data were not available.
  Carbon dioxide; intolerance Day6; n= 0,0,2,1,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.50 (NA) — NA indicates that data were not available. | 5.00 (NA) — NA indicates that data were not available. | 2.00 (NA) — NA indicates that data were not available. | 4.15 (NA) — NA indicates that data were not available.
  Carbon dioxide; intolerance Day7; n= 0,0,1,0,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.00 (NA) — NA indicates that data were not available. | 2.65 (NA) — NA indicates that data were not available.
  Carbon dioxide; follow up; n= 15,20,3,3,3,2 | -1.26 (6.069) | -0.40 (5.088) | 1.67 (2.082) | 1.67 (3.215) | 1.67 (1.528) | 1.45 (NA) — NA indicates that data were not available.
  Glucose; Day2; n= 31,35,2,2,0,0 | 0.2871 (2.68325) | -0.2338 (1.89890) | -0.8000 (NA) — NA indicates that data were not available. | 0.3000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Glucose; Day3; n= 29,29,1,1,0,0 | 0.2414 (3.12667) | 0.0655 (2.10514) | -2.9000 (NA) — NA indicates that data were not available. | -1.6000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Glucose; Day4; n= 25,24,0,0,0,0 | 0.7680 (2.69764) | -0.1458 (1.96778) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Glucose; Day5; n= 22,21,0,0,0,0 | 0.4636 (2.76811) | 0.1810 (2.05928) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Glucose; Day6; n= 18,18,0,0,0,0 | 0.8111 (3.37445) | 0.0889 (1.74150) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Glucose; Day7; n= 14,13,0,0,0,0 | 1.8857 (4.17702) | 0.8692 (2.33323) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Glucose; intolerance Day1; n= 1,0,2,3,0,0 | -0.9000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.6000 (NA) — NA indicates that data were not available. | -0.2000 (1.30000) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Glucose; intolerance Day2; n= 0,0,3,3,4,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.5000 (2.85132) | -0.3000 (0.62450) | -0.4500 (2.49600) | 0.8000 (1.50000)
  Glucose; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.5000 (NA) — NA indicates that data were not available. | 0.1000 (1.21244) | 0.7333 (1.90875) | 0.6000 (1.78699)
  Glucose; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.8500 (NA) — NA indicates that data were not available. | -0.3000 (NA) — NA indicates that data were not available. | 2.1000 (2.88444) | 1.1667 (0.32146)
  Glucose; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.5500 (NA) — NA indicates that data were not available. | 0.2000 (NA) — NA indicates that data were not available. | 1.2333 (3.27159) | 0.9333 (0.87369)
  Glucose; intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.1000 (NA) — NA indicates that data were not available. | -0.7000 (NA) — NA indicates that data were not available. | 0.8000 (1.70880) | 0.6500 (NA) — NA indicates that data were not available.
  Glucose; intolerance Day7; n= 0,0,1,0,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.8000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 2.5000 (NA) — NA indicates that data were not available. | 0.1500 (NA) — NA indicates that data were not available.
  Glucose; follow up; n= 18,17,3,3,4,2 | -0.8889 (2.55225) | -1.7176 (1.99663) | -1.9667 (3.21921) | -0.3333 (0.72342) | -1.1750 (2.57083) | 2.6000 (NA) — NA indicates that data were not available.
  Potassium; Day2; n= 33,37,2,2,0,0 | -0.08 (0.474) | 0.02 (0.447) | -0.20 (NA) — NA indicates that data were not available. | -0.20 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Potassium; Day3; n= 29,31,1,1,0,0 | -0.12 (0.582) | 0.01 (0.489) | -0.40 (NA) — NA indicates that data were not available. | -0.10 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Potassium; DAY4; n= 24,25,0,0,0,0 | 0.08 (0.705) | 0.06 (0.515) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Potassium Day5; n= 22,23,0,0,0,0 | 0.10 (0.559) | 0.07 (0.644) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Potassium; Day6; n= 18,19,0,0,0,0 | 0.33 (0.428) | 0.09 (0.732) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Potassium; Day7; n= 14,15,0,0,0,0 | 0.49 (0.350) | 0.05 (0.741) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Potassium; intolerance Day1; n= 1,0,2,3,0,0 | 0.40 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.00 (NA) — NA indicates that data were not available. | 0.17 (0.379) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Potassium; intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.00 (0.557) | 0.17 (0.289) | 0.40 (0.258) | -0.18 (0.263)
  Potassium; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.30 (NA) — NA indicates that data were not available. | 0.30 (0.656) | 0.30 (0.721) | -0.53 (1.011)
  Potassium; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.15 (NA) — NA indicates that data were not available. | 0.45 (NA) — NA indicates that data were not available. | 0.63 (0.945) | -0.10 (1.136)
  Potassium; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.35 (NA) — NA indicates that data were not available. | 0.20 (NA) — NA indicates that data were not available. | 0.67 (0.987) | -0.03 (1.115)
  Potassium; intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.05 (NA) — NA indicates that data were not available. | 0.40 (NA) — NA indicates that data were not available. | 0.83 (1.115) | -0.55 (NA) — NA indicates that data were not available.
  Potassium; intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.10 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.87 (1.328) | -0.60 (NA) — NA indicates that data were not available.
  Potassium; follow up; n= 25,28,3,3,4,2 | 0.37 (0.471) | 0.11 (0.676) | -0.07 (0.379) | 0.47 (0.651) | 0.38 (0.443) | -0.10 (NA) — NA indicates that data were not available.
  Sodium; Day2; n= 33,37,2,2,0,0 | 0.3 (2.02) | 0.8 (3.34) | 1.5 (NA) — NA indicates that data were not available. | -0.5 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Sodium; Day3; n= 29,31,1,1,0,0 | 0.4 (2.47) | 1.2 (4.20) | 0.0 (NA) — NA indicates that data were not available. | -5.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Sodium; Day4; n= 25,26,0,0,0,0 | -0.8 (4.03) | 1.5 (4.92) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Sodium; Day5; n= 22,23,0,0,0,0 | -1.4 (4.62) | 0.8 (5.24) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Sodium; Day6; n= 18,19,0,0,0,0 | -2.8 (6.18) | -0.2 (6.39) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Sodium; Day7; n= 14,15,0,0,0,0 | -2.7 (6.40) | 0.1 (4.24) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Sodium; intolerance Day1; n= 1,0,2,3,0,0 | -3.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.5 (NA) — NA indicates that data were not available. | -2.3 (6.66) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Sodium; intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0 (2.65) | -3.3 (6.66) | -0.5 (2.38) | 1.0 (2.16)
  Sodium; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.5 (NA) — NA indicates that data were not available. | -3.0 (8.89) | 3.7 (3.21) | -0.5 (4.65)
  Sodium; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 2.0 (NA) — NA indicates that data were not available. | -8.0 (NA) — NA indicates that data were not available. | 3.7 (2.31) | 0.0 (6.93)
  Sodium; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 5.0 (NA) — NA indicates that data were not available. | 1.0 (NA) — NA indicates that data were not available. | 6.3 (2.31) | 0.0 (6.08)
  Sodium; intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.5 (NA) — NA indicates that data were not available. | -2.0 (NA) — NA indicates that data were not available. | 7.3 (2.52) | -1.0 (NA) — NA indicates that data were not available.
  Sodium; intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 2.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 6.3 (6.66) | -2.5 (NA) — NA indicates that data were not available.
  Sodium; follow up; n= 25,28,3,3,4,2 | -3.8 (4.92) | -2.5 (5.12) | -3.0 (3.46) | -7.0 (6.08) | -0.5 (5.45) | -6.5 (NA) — NA indicates that data were not available.
  BUN; Day2; n= 1,3,0,0,0,0 | 1.0000 (NA) — NA indicates that data were not available. | 2.3000 (4.60326) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; Day3; n= 1,2,0,0,0,0 | 6.4000 (NA) — NA indicates that data were not available. | 2.4000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; Day4; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 1.5000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; Day5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 25.8500 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; Day6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 29.2000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; Day7; n= 13,14,0,0,0,0 | 3.1231 (5.15948) | 5.0143 (9.35002) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; intolerance Day3; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.2000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; intolerance Day4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.3000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; intolerance Day6; n= 0,0,1,1,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 7.4000 (NA) — NA indicates that data were not available. | 2.2000 (NA) — NA indicates that data were not available. | 14.2000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  BUN; intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.0000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 16.4000 (18.72004) | 1.1500 (NA) — NA indicates that data were not available.
  BUN; follow up; n= 18,22,3,3,4,1 | 2.1722 (5.48397) | 1.7000 (6.75891) | -0.3333 (3.30807) | 4.5667 (1.59478) | 11.6500 (21.03656) | 2.8000 (NA) — NA indicates that data were not available.

14. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet and White Blood Cell (WBC) Levels
Description: Blood samples were collected to evaluate change from Baseline in basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet and WBC values at Baseline up to Day 7 and follow up (till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Giga unit per liter (gI/L)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
Giga unit per liter (gI/L)
  Basophils; Day2; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Basophils; Day3; n= 2,1,0,0,0,0 | 0.000 (NA) — NA indicates that data were not available. | -0.020 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Basophils; Day5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.050 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Basophils; Day6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Basophils; Day7; n= 13,14,0,0,0,0 | 0.022 (0.0402) | 0.013 (0.0281) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Basophils; intolerance Day2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — c | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.030 (NA) — NA indicates that data were not available.
  Basophils; intolerance Day3; n= 0,0,0,2,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Basophils; intolerance Day4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Basophils; intolerance Day6; n= 0,0,1,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.000 (NA) — NA indicates that data were not available. | 0.020 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Basophils; intolerance Day7; n= 0,0,1,0,3,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.130 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.037 (0.0603) | 0.300 (NA) — NA indicates that data were not available.
  Basophils; follow up; n= 24,28,3,3,3,1 | 0.040 (0.0546) | 0.034 (0.0619) | 0.047 (0.0503) | 0.057 (0.0379) | 0.073 (0.1401) | 0.150 (NA) — NA indicates that data were not available.
  Eosinophils; Day2; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.0000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Eosinophils; Day3; n= 2,1,0,0,0,0 | 0.3000 (NA) — NA indicates that data were not available. | -0.0400 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Eosinophils; Day5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.0900 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Eosinophils; Day6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.2000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Eosinophils; Day7; n= 13,14,0,0,0,0 | 0.1615 (0.12877) | 0.1079 (0.22337) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Eosinophils; intolerance Day2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.0200 (NA) — NA indicates that data were not available.
  Eosinophils; intolerance Day3; n= 0,0,0,2,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0300 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Eosinophils; intolerance Day4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Eosinophils; intolerance Day6; n= 0,0,1,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0000 (NA) — NA indicates that data were not available. | 0.3300 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Eosinophils; intolerance Day7; n= 0,0,1,0,3,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.7900 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.0000 (0.19079) | 0.1000 (NA) — NA indicates that data were not available.
  Eosinophils; follow up; n= 24,28,3,3,4,1 | 1.4454 (6.27749) | 0.1886 (0.27639) | 0.3367 (0.14844) | 0.2267 (0.14189) | 0.0400 (0.81404) | -0.0200 (NA) — NA indicates that data were not available.
  Lymphocytes; Day2; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.2000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Lymphocytes; Day3; n= 2,1,0,0,0,0 | 0.6500 (NA) — NA indicates that data were not available. | -1.0300 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Lymphocytes; Day5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.4400 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Lymphocytes; Day6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.2000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Lymphocytes; Day7; n= 13,15,0,0,0,0 | 0.3946 (0.56592) | 0.2320 (0.66890) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Lymphocytes; intolerance Day2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.7300 (NA) — NA indicates that data were not available.
  Lymphocytes; intolerance Day3; n= 0,0,0,2,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.3550 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Lymphocytes; intolerance Day4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.2000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Lymphocytes; intolerance Day6; n= 0,0,1,1,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.1000 (NA) — NA indicates that data were not available. | 0.4800 (NA) — NA indicates that data were not available. | 0.4000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Lymphocytes; intolerance Day7; n= 0,0,1,0,3,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.4600 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.1900 (0.19925) | 1.5000 (NA) — NA indicates that data were not available.
  Lymphocytes; follow up; n= 24,28,3,3,4,2 | 0.6483 (0.51967) | 0.6614 (0.75393) | 0.3133 (0.53529) | 0.7067 (0.50013) | 0.7100 (0.58395) | -0.1200 (NA) — NA indicates that data were not available.
  Monocytes; Day2; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.4000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Monocytes; Day3; n= 2,1,0,0,0,0 | 0.5000 (NA) — NA indicates that data were not available. | -0.0600 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Monocytes; Day5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.0300 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Monocytes; Day6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.2000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Monocytes; Day7; n= 13,15,0,0,0,0 | 0.2100 (0.59020) | 0.1647 (0.49461) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Monocytes; intolerance Day2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0600 (NA) — NA indicates that data were not available.
  Monocytes; intolerance Day3; n= 0,0,0,2,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0900 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Monocytes; intolerance Day4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.1000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Monocytes; intolerance Day6; n= 0,0,1,1,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.9000 (NA) — NA indicates that data were not available. | 0.3600 (NA) — NA indicates that data were not available. | 0.5000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Monocytes; intolerance Day7; n= 0,0,1,0,3,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.6900 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0600 (0.29866) | 1.3000 (NA) — NA indicates that data were not available.
  Monocytes; follow up; n= 24,28,3,3,3,1 | 0.1475 (0.55989) | 0.0611 (0.39000) | -0.1067 (0.46058) | -0.0633 (0.20502) | -0.4900 (0.56427) | 0.3600 (NA) — NA indicates that data were not available.
  Neutrophils; Day2; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -1.5000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Neutrophils; Day3; n= 2,1,0,0,0,0 | -5.3000 (NA) — NA indicates that data were not available. | 0.7200 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Neutrophils; Day5; n= 0,2,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.3750 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Neutrophils; Day6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 9.6000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Neutrophils; Day7; n= 13,15,0,0,0,0 | 0.6708 (7.11859) | 1.1807 (3.99306) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Neutrophils; intolerance Day2; n= 0,0,0,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.3100 (NA) — NA indicates that data were not available.
  Neutrophils; intolerance Day3; n= 0,0,0,2,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -2.1000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Neutrophils; intolerance Day4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -2.9000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Neutrophils; intolerance Day6; n= 0,0,1,1,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.1000 (NA) — NA indicates that data were not available. | -0.8100 (NA) — NA indicates that data were not available. | 7.5000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Neutrophils; intolerance Day7; n= 0,0,1,0,3,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.4600 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.7200 (8.10489) | -6.6000 (NA) — NA indicates that data were not available.
  Neutrophils; follow up; n= 24,28,3,3,4,2 | -2.0579 (6.73610) | -2.0968 (3.26061) | -0.7133 (5.15272) | -0.5233 (1.90500) | 0.8250 (12.60760) | -6.7400 (NA) — NA indicates that data were not available.
  Platelet; Day2; n= 32,37,2,2,0,0 | 10.5 (40.92) | 4.2 (22.00) | 8.5 (NA) — NA indicates that data were not available. | 14.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Platelet; Day3; n= 29,30,1,1,0,0 | 34.8 (65.68) | 22.1 (35.90) | -4.0 (NA) — NA indicates that data were not available. | 10.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Platelet; Day4; n= 25,26,0,0,0,0 | 56.0 (98.65) | 48.7 (55.92) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Platelet; Day5; n= 22,23,0,0,0,0 | 102.7 (141.00) | 82.7 (75.37) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Platelet; Day6; n= 17,19,0,0,0,0 | 128.7 (168.94) | 113.6 (95.44) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Platelet; Day7; n= 14,15,0,0,0,0 | 159.8 (229.46) | 133.3 (99.92) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Platelet; intolerance Day1; n= 1,0,2,3,0,0 | -24.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 33.5 (NA) — NA indicates that data were not available. | 21.0 (39.89) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Platelet; intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 73.7 (21.20) | 13.7 (73.15) | -8.8 (24.25) | 16.3 (30.10)
  Platelet; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 101.5 (NA) — NA indicates that data were not available. | 31.7 (64.79) | 0.7 (46.70) | 29.0 (56.94)
  Platelet; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 183.0 (NA) — NA indicates that data were not available. | 42.5 (NA) — NA indicates that data were not available. | 11.0 (67.58) | 86.3 (57.36)
  Platelet; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 213.5 (NA) — NA indicates that data were not available. | -10.0 (NA) — NA indicates that data were not available. | 14.7 (75.24) | 158.0 (99.05)
  Platelet; intolerance day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 225.5 (NA) — NA indicates that data were not available. | 42.0 (NA) — NA indicates that data were not available. | 26.0 (84.55) | 271.0 (NA) — NA indicates that data were not available.
  Platelet; intolerance day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 287.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 49.7 (106.59) | 429.0 (NA) — NA indicates that data were not available.
  Platelet; follow up; n= 24,28,3,3,4,2 | 258.9 (268.60) | 272.0 (226.86) | 438.0 (194.76) | 272.0 (27.87) | 66.8 (272.20) | 891.0 (NA) — NA indicates that data were not available.
  WBC; Day2; n= 32,37,2,2,0,0 | -1.187 (3.5946) | -0.199 (2.5427) | -2.490 (NA) — NA indicates that data were not available. | -2.320 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  WBC; Day3; n= 29,30,1,1,0,0 | -1.033 (5.8272) | 0.398 (3.0461) | 0.300 (NA) — NA indicates that data were not available. | -4.400 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  WBC; Day4; n= 25,26,0,0,0,0 | -1.398 (6.0244) | 0.489 (3.7565) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  WBC; Day5; n= 22,23,0,0,0,0 | -0.015 (6.5214) | 1.320 (3.6270) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  WBC; Day6; n= 17,19,0,0,0,0 | 0.881 (8.4975) | 2.314 (4.6829) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  WBC; Day7; n= 14,15,0,0,0,0 | 0.690 (8.9417) | 1.913 (3.8002) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  WBC; intolerance Day1; n= 1,0,2,3,0,0 | -2.020 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.300 (NA) — NA indicates that data were not available. | -1.220 (2.6018) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  WBC; intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.197 (2.1019) | -1.713 (3.4082) | -1.050 (3.3491) | 0.450 (4.6177)
  WBC; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.910 (NA) — NA indicates that data were not available. | -1.447 (2.4791) | -2.333 (5.1733) | -2.925 (4.9304)
  WBC; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.150 (NA) — NA indicates that data were not available. | -2.125 (NA) — NA indicates that data were not available. | -1.300 (4.8446) | -2.933 (6.4733)
  WBC; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.850 (NA) — NA indicates that data were not available. | -0.490 (NA) — NA indicates that data were not available. | -1.450 (8.5339) | -1.800 (5.4009)
  WBC; intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.750 (NA) — NA indicates that data were not available. | 0.300 (NA) — NA indicates that data were not available. | -0.367 (8.8047) | -5.600 (NA) — NA indicates that data were not available.
  WBC; intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.000 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.540 (8.7199) | -3.650 (NA) — NA indicates that data were not available.
  WBC; follow up; n= 24,28,3,3,4,2 | -1.223 (7.5546) | -0.813 (3.7488) | -0.177 (5.0906) | 0.230 (2.4557) | 2.188 (13.4717) | -6.150 (NA) — NA indicates that data were not available.

15. Secondary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) Levels
Description: Blood samples were collected to evaluate change from Baseline in hemoglobin and MCHC values at Baseline up to Day 7 and follow up (till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
g/L
  Hemoglobin; Day2; n= 32,37,2,2,0,0 | -2.7 (8.13) | -1.8 (6.62) | -10.5 (NA) — NA indicates that data were not available. | -4.5 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Hemoglobin; Day3; n= 29,30,1,1,0,0 | -4.6 (8.91) | -2.1 (8.67) | -6.0 (NA) — NA indicates that data were not available. | -7.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Hemoglobin; Day4; n= 25,26,0,0,0,0 | -4.8 (7.71) | -4.7 (7.59) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Hemoglobin; Day5; n= 22,23,0,0,0,0 | -3.2 (10.40) | -3.6 (10.28) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Hemoglobin; Day6; n= 17,19,0,0,0,0 | -5.6 (14.04) | -4.7 (10.19) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Hemoglobin; Day7; n= 14,15,0,0,0,0 | -5.9 (14.22) | -5.9 (11.06) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Hemoglobin; Intolerance Day1; n= 1,0,2,3,0,0 | -16.0 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 2.0 (NA) — NA indicates that data were not available. | -4.0 (1.73) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Hemoglobin; Intolerance Day2; n= 0,0,3,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -4.7 (3.06) | -8.7 (7.57) | 0.5 (4.20) | -4.5 (2.52)
  Hemoglobin; Intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -11.5 (NA) — NA indicates that data were not available | -11.0 (4.58) | -2.7 (7.09) | -3.8 (4.27)
  Hemoglobin; Intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -5.0 (NA) — NA indicates that data were not available | -10.0 (NA) — NA indicates that data were not available | -0.7 (8.74) | -1.7 (5.69)
  Hemoglobin; Intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -13.0 (NA) — NA indicates that data were not available | -6.0 (NA) — NA indicates that data were not available | -7.0 (10.00) | 4.3 (1.53)
  Hemoglobin; Intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -14.0 (NA) — NA indicates that data were not available | -7.0 (NA) — NA indicates that data were not available | 5.7 (10.02) | -5.5 (NA) — NA indicates that data were not available
  Hemoglobin; Intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -13.0 (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | 2.7 (9.24) | -5.5 (NA) — NA indicates that data were not available
  Hemoglobin; follow up; n= 24,28,3,3,4,2 | 5.1 (19.13) | 4.3 (13.21) | 15.7 (9.87) | 19.0 (8.19) | 3.5 (8.81) | 2.5 (NA) — NA indicates that data were not available
  MCHC; Day2; n= 31,37,2,2,0,0 | -1.26 (7.066) | -0.27 (5.966) | -2.50 (NA) — NA indicates that data were not available | 3.00 (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available
  MCHC; Day3; n= 28,30,1,1,0,0 | -1.29 (7.403) | -2.00 (7.339) | -13.00 (NA) — NA indicates that data were not available | 6.00 (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available
  MCHC; Day4; n= 25,26,0,0,0,0 | -1.24 (8.232) | -5.54 (8.994) | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available
  MCHC; Day5; n= 22,23,0,0,0,0 | -16.50 (68.162) | -6.39 (9.852) | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available
  MCHC; Day6; n= 17,19,0,0,0,0 | -1.94 (10.413) | -6.89 (11.110) | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available
  MCHC; Day7; n= 14,15,0,0,0,0 | -4.43 (13.461) | -4.40 (9.934) | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available
  MCHC; intolerance Day1; n= 1,0,2,3,0,0 | 0.00 (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -18.50 (NA) — NA indicates that data were not available | 1.00 (8.544) | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available
  MCHC; intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -19.00 (23.065) | 1.67 (12.702) | -0.50 (4.655) | -3.00 (6.831)
  MCHC; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -6.00 (NA) — NA indicates that data were not available | 5.33 (9.609) | -2.67 (9.815) | -3.75 (11.325)
  MCHC; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -12.50 (NA) — NA indicates that data were not available | 2.00 (NA) — NA indicates that data were not available | -4.00 (6.557) | -11.67 (18.230)
  MCHC; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -6.50 (NA) — NA indicates that data were not available | -5.00 (NA) — NA indicates that data were not available | -10.00 (12.288) | -11.67 (23.352)
  MCHC; intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -13.00 (NA) — NA indicates that data were not available | -10.00 (NA) — NA indicates that data were not available | -8.00 (18.248) | -23.50 (NA) — NA indicates that data were not available
  MCHC; intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -25.00 (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available | -8.67 (15.535) | -8.50 (NA) — NA indicates that data were not available
  MCHC; follow up; n= 23,27,3,3,4,4 | -2.57 (10.135) | -6.33 (14.475) | -22.00 (29.138) | -5.33 (9.609) | -11.75 (11.026) | -25.00 (NA) — NA indicates that data were not available

16. Secondary Outcome: Change From Baseline in Hematocrit Level
Description: Blood samples were collected to evaluate change from Baseline in hematocrit values at Baseline up to Day 7 and follow up (till day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Fraction of 1
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
Fraction of 1
  Day2; n= 32,37,2,2,0,0 | -0.0072 (0.02369) | -0.0048 (0.02013) | -0.0310 (NA) — NA indicates that the data was not available | -0.0195 (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available
  Day3; n= 29,30,1,1,0,0 | -0.0129 (0.02555) | -0.0046 (0.02342) | -0.0090 (NA) — NA indicates that the data was not available | -0.0300 (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available
  Day4; n= 25,26,0,0,0,0 | -0.0140 (0.02358) | -0.0107 (0.02226) | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available
  Day5; n= 22,23,0,0,0,0 | -0.0085 (0.02886) | -0.0064 (0.02956) | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available
  Day6; n= 17,19,0,0,0,0 | -0.0152 (0.03950) | -0.0088 (0.03036) | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available
  Day7; n= 14,15,0,0,0,0 | -0.0148 (0.04008) | -0.0145 (0.03551) | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available
  Intolerance Day1; n= 1,0,2,3,0,0 | -0.0400 (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | 0.0195 (NA) — NA indicates that the data was not available | -0.0150 (0.00500) | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available
  Intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | -0.0017 (0.02438) | -0.0287 (0.02203) | -0.1385 (0.26790) | -0.0113 (0.00699)
  Intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | -0.0310 (NA) — NA indicates that the data was not available | -0.0373 (0.02053) | -0.1917 (0.30168) | -0.0065 (0.00790)
  Intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | -0.0050 (NA) — NA indicates that the data was not available | -0.0350 (NA) — NA indicates that the data was not available | -0.1803 (0.29416) | 0.0030 (0.01836)
  Intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | -0.0350 (NA) — NA indicates that the data was not available | -0.0200 (NA) — NA indicates that the data was not available | -0.1963 (0.29767) | 0.0213 (0.01474)
  Intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | -0.0320 (NA) — NA indicates that the data was not available | -0.0200 (NA) — NA indicates that the data was not available | -0.1617 (0.30168) | -0.0030 (NA) — NA indicates that the data was not available
  Intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | -0.0200 (NA) — NA indicates that the data was not available | NA (NA) — NA indicates that the data was not available | -0.1673 (0.31439) | -0.0120 (NA) — NA indicates that the data was not available
  Follow up; n= 24,28,3,3,4,2 | 0.0183 (0.05406) | 0.0179 (0.04098) | 0.0650 (0.05679) | 0.0607 (0.01793) | -0.1180 (0.26962) | 0.0320 (NA) — NA indicates that the data was not available

17. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV) Levels
Description: Blood samples were collected to evaluate change from Baseline in MCV values at Baseline up to Day 7 and follow up (till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
Femtoliter (fL)
  Day2; n= 31,37,2,2,0,0 | 0.36 (1.349) | 0.14 (1.478) | 1.70 (NA) — NA indicates that data were not available. | -0.50 (NA) — NA indicates that data were not available. | -0.60 (0.876) | NA (NA) — NA indicates that data were not available.
  Day3; n= 28,30,1,1,0,0 | 0.13 (1.431) | 0.40 (1.627) | 3.90 (NA) — NA indicates that data were not available. | 0.00 (NA) — NA indicates that data were not available. | -2.47 (3.101) | NA (NA) — NA indicates that data were not available.
  Day4; n= 25,26,0,0,0,0 | -0.14 (2.108) | 0.79 (2.017) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -2.53 (2.194) | NA (NA) — NA indicates that data were not available.
  Day5; n= 22,23,0,0,0,0 | 0.09 (2.661) | 0.40 (2.042) | NA (NA) — NA indicates that data were not available | NA (NA) — NA indicates that data were not available. | -1.10 (3.804) | NA (NA) — NA indicates that data were not available.
  Day6; n= 17,19,0,0,0,0 | 0.17 (3.098) | 0.53 (2.515) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -2.20 (5.800) | NA (NA) — NA indicates that data were not available.
  Day7; n= 14,15,0,0,0,0 | 1.04 (3.680) | -0.01 (2.669) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -1.13 (5.244) | NA (NA) — NA indicates that data were not available.
  Intolerance Day1; n= 1,0,2,3,0,0 | 0.50 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.10 (NA) — NA indicates that data were not available. | -1.10 (0.854) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.43 (3.182) | 0.00 (1.732) | NA (NA) — NA indicates that data were not available. | 0.92 (1.187)
  Intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 1.30 (NA) — NA indicates that data were not available. | -1.20 (1.709) | NA (NA) — NA indicates that data were not available. | 0.27 (2.968)
  Intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.05 (NA) — NA indicates that data were not available. | -1.10 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 2.30 (4.107)
  Intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 2.90 (NA) — NA indicates that data were not available. | 0.10 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.13 (5.169)
  Intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 3.95 (NA) — NA indicates that data were not available. | -0.20 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 5.60 (NA) — NA indicates that data were not available.
  Intolerance Day7; n= 0,01,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 5.10 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 4.15 (NA) — NA indicates that data were not available.
  Follow up; n= 23,27,3,3,4,2 | -0.24 (3.394) | 1.46 (4.280) | 4.57 (3.774) | -2.93 (0.902) | -0.77 (5.557) | 4.00 (NA) — NA indicates that data were not available.

18. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) and Reticulocyte Count
Description: Blood samples were collected to evaluate change from Baseline in RBC and reticulocytes values at Baseline up to Day 7 and follow up (till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Tetra unit per liter (TI/L)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
Tetra unit per liter (TI/L)
  RBC; Day2; n= 32,37,2,2,0,0 | -0.098 (0.2816) | -0.059 (0.2262) | -0.375 (NA) — NA indicates that data were not available. | -0.150 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  RBC; Day3; n= 29,30,1,1,0,0 | -0.163 (0.3001) | -0.067 (0.2776) | -0.210 (NA) — NA indicates that data were not available. | -0.200 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  RBC; Day4; n= 25,26,0,0,0,0 | -0.155 (0.3038) | -0.141 (0.2417) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  RBC; Day5; n= 22,23,0,0,0,0 | -0.099 (0.3676) | -0.085 (0.3246) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  RBC; Day6; n= 17,19,0,0,0,0 | -0.176 (0.4999) | -0.118 (0.3403) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  RBC; Day7; n= 14,15,0,0,0,0 | -0.202 (0.4849) | -0.149 (0.3610) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  RBC; intolerance Day1; n= 1,0,2,3,0,0 | -0.540 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.120 (NA) — NA indicates that data were not available. | -0.077 (0.0586) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  RBC; intolerance Day2; n= 0,0,3,3,4,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.113 (0.1701) | -0.293 (0.2335) | 0.018 (0.1228) | -0.172 (0.1159)
  RBC; intolerance Day3; n= 0,0,2,3,3,4 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.390 (NA) — NA indicates that data were not available. | -0.333 (0.1563) | -0.030 (0.2042) | -0.105 (0.1511)
  RBC; intolerance Day4; n= 0,0,2,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.165 (NA) — NA indicates that data were not available. | -0.270 (NA) — NA indicates that data were not available. | 0.047 (0.3075) | -0.050 (0.2390)
  RBC; intolerance Day5; n= 0,0,2,1,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.495 (NA) — NA indicates that data were not available. | -0.150 (NA) — NA indicates that data were not available. | -0.157 (0.3371) | 0.133 (0.0306)
  RBC; intolerance Day6; n= 0,0,2,1,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.505 (NA) — NA indicates that data were not available. | -0.130 (NA) — NA indicates that data were not available. | 0.267 (0.3055) | -0.170 (NA) — NA indicates that data were not available.
  RBC; intolerance Day7; n= 0,0,1,0,3,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.400 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.150 (0.2598) | -0.250 (NA) — NA indicates that data were not available.
  RBC follow up; n= 24,28,3,3,4,2 | 0.195 (0.6553) | 0.142 (0.4196) | 0.577 (0.4826) | 0.790 (0.1493) | 0.188 (0.3636) | 0.170 (NA) — NA indicates that data were not available.
  Reticulocytes; Day5; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | -0.0010 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Reticulocytes; Day6; n= 0,1,0,0,0,0 | NA (NA) — NA indicates that data were not available. | 0.0810 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Reticulocytes; Day7; n= 7,4,0,0,0,0 | 0.0074 (0.04599) | 0.0031 (0.01158) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Reticulocytes; intolerance Day3; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0530 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Reticulocytes; intolerance Day4; n= 0,0,0,1,0,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0080 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Reticulocytes; intolerance Day6; n= 0,0,0,0,1,0 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0340 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Reticulocytes; intolerance Day7; n= 0,0,1,0,0,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0170 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.0822 (NA) — NA indicates that data were not available.
  Reticulocytes; follow up; n= 11,11,2,2,3,2 | 4.1273 (13.55607) | 1.6622 (5.41884) | 0.0847 (NA) — NA indicates that data were not available. | 0.0537 (NA) — NA indicates that data were not available. | 0.0870 (0.02364) | 0.0569 (NA) — NA indicates that data were not available.

19. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) Levels
Description: Blood samples were collected to evaluate change from Baseline in MCH values at Baseline up to Day 7 and follow up (till Day 23). Blood samples were also collected on Day 9 for those participants who completed 7 days of dosing. Change from Baseline was defined as post dose visit value minus Baseline value. For participants who developed intolerance, blood samples were taken for Day 1 to Day 7 up to 6 hrs prior to dosing. NA indicates that data were not available. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). If n < 3 the SD was set to missing.
Time Frame: Up to 23 days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picogram (PG)
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Number analyzed (Participants) | 35 | 39 | 3 | 3 | 4 | 4
Picogram (PG)
  Day2; n= 27,35,2,1,0,0 | 0.01 (0.522) | 0.02 (0.531) | 0.35 (NA) — NA indicates that data were not available. | 0.00 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Day3; n= 24,28,1,0,0,0 | -0.10 (0.581) | -0.08 (0.547) | 0.20 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Day4; n= 21,24,0,0,0,0 | -0.26 (0.685) | -0.24 (0.690) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Day5; n= 19,21,0,0,0,0 | -0.23 (0.628) | -0.44 (0.494) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Day6; n= 15,17,0,0,0,0 | -0.15 (0.505) | -0.41 (0.431) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Day7; n= 12,14,0,0,0,0 | -0.02 (0.488) | -0.45 (0.435) | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Intolerance Day1; n= 1,0,2,2,0,0 | 0.20 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.65 (NA) — NA indicates that data were not available. | -0.30 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available.
  Intolerance Day2; n= 0,0,3,2,3,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.57 (1.060) | -0.10 (NA) — NA indicates that data were not available. | -0.23 (0.681) | -0.10 (0.265)
  Intolerance Day3; n= 0,0,2,2,2,3 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.10 (NA) — NA indicates that data were not available. | -0.10 (NA) — NA indicates that data were not available. | -0.65 (NA) — NA indicates that data were not available. | -0.27 (0.153)
  Intolerance Day4; n= 0,0,2,1,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.10 (NA) — NA indicates that data were not available. | -0.60 (NA) — NA indicates that data were not available. | -0.75 (NA) — NA indicates that data were not available. | -0.50 (NA) — NA indicates that data were not available.
  Intolerance Day5; n= 0,0,2,1,2,2 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.45 (NA) — NA indicates that data were not available. | -0.50 (NA) — NA indicates that data were not available. | -1.00 (NA) — NA indicates that data were not available. | -0.30 (NA) — NA indicates that data were not available.
  Intolerance Day6; n= 0,0,2,1,2,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | 0.20 (NA) — NA indicates that data were not available. | -1.10 (NA) — NA indicates that data were not available. | -1.00 (NA) — NA indicates that data were not available. | -0.70 (NA) — NA indicates that data were not available.
  Intolerance Day7; n= 0,0,1,0,2,1 | NA (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.50 (NA) — NA indicates that data were not available. | NA (NA) — NA indicates that data were not available. | -0.75 (NA) — NA indicates that data were not available. | 0.40 (NA) — NA indicates that data were not available.
  Follow up; n= 21,26,3,2,3,2 | -0.40 (0.889) | -0.20 (0.944) | -0.50 (1.652) | -2.15 (NA) — NA indicates that data were not available. | -0.50 (0.800) | -0.90 (NA) — NA indicates that data were not available.

20. Secondary Outcome: Log Transformed Concentration at 60 Minutes (Min) (C60) and Maximum Observed Concentration (Cmax) of Acetaminophen (Prior to Intolerance)
Description: Blood samples for pharmacokinetic (PK) analysis were collected at Baseline, and at Day 2 or at Day 3 (OR very rarely Day 4 - only if Day 2 or Day 3 sample could not be obtained) prior to intolerance. Prior to intolerance was defined as prior to development of intolerance. C60 was defined as observed plasma concentration at 60 min after administration of enteral feed with acetaminophen and Cmax was defined as maximum observed plasma concentration of acetaminophen. The absorption profile of acetaminophen was used as an indirect measure of gastric emptying function. The analysis was performed on ITT (exposed) Population. Due to change in sampling schedule, samples were only obtained to 4 hours. Only those participants available at the specified time points were analyzed (represented by n= x in the category titles).
Time Frame: At Day 2
Population: ITT (exposed) Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Log [nanogram per milliliter (ng/mL)]
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
Log [nanogram per milliliter (ng/mL)]
  C60; Pre-dose; n= 42,36 | 4108.99 [3357.46 to 5028.74] | 4374.35 [3157.08 to 6060.97]
  C60; post-dose; n= 33,27 | 4504.30 [3428.13 to 5918.29] | 4691.64 [3917.56 to 5618.66]
  Cmax; pre-dose; n= 42,36 | 5482.09 [4529.01 to 6635.72] | 6068.34 [4428.15 to 8316.07]
  Cmax; post-dose; n= 33,27 | 6576.47 [5123.54 to 8441.42] | 6319.73 [5251.08 to 7605.87]

21. Secondary Outcome: Log Transformed AUC[0-60] of Acetaminophen
Description: Blood samples for PK analysis were collected at Baseline, and at 60 min. at Day 2 or Day 3 (or very rarely Day 4 - only if Day 2 or Day 3 sample could not be obtained) prior to intolerance. Prior to intolerance was defined as prior to development of intolerance. AUC[0-60] of acetaminophen was defined as area under the concentration-time curve from time zero to 60 min. and it was calculated as Log trapezoidal rule from concentration-time data. The absorption profile of acetaminophen was used as an indirect measure of gastric emptying function. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles)
Time Frame: At Day 2
Population: ITT (exposed) Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Log [min into ng/mL (min*ng/mL)]
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
Log [min into ng/mL (min*ng/mL)]
  Pre-dose; n=42,36 | 192321.7 [153049.5 to 241671.0] | 222411.3 [161086.4 to 307082.4]
  Post-dose; n= 33,27 | 234538.9 [174645.6 to 314972.3] | 228473.7 [185338.9 to 281647.5]

22. Secondary Outcome: Log Transformed AUC[0-60] of 3-O-methylglucose (3- OMG)
Description: Blood samples for PK analysis were collected at Baseline, and at Day 2 or Day 3 (or very rarely Day 4 - only if Day 2 or Day 3 sample could not be obtained) prior to intolerance. Prior to intolerance was defined as prior to development of intolerance. AUC[0-60] of 3-OMG was defined as area under the concentration-time curve from time zero to 60 min. and it was calculated as Log trapezoidal rule from concentration-time data. The absorption profile of 3-OMG was used as an indirect measure of gastric emptying function. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles)
Time Frame: At Day 2
Population: ITT (exposed) Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Log [Min. into mmol/L (min*mmol/l)]
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
Log [Min. into mmol/L (min*mmol/l)]
  Pre-dose; n=38,34 | 3.3709 [2.2283 to 5.0993] | 3.8341 [2.5286 to 5.8136]
  Post-dose; n= 32,27 | 7.2872 [5.9044 to 8.9938] | 6.1047 [4.3137 to 8.6394]

23. Secondary Outcome: Log Transformed C60 of 3-OMG
Description: Blood samples for PK analysis were collected at Baseline and at Day 2 or Day 3 (or very rarely at Day 4 - only if Day 2 or Day 3 sample could not be obtained)prior to intolerance. Prior to intolerance was defined as prior to development of intolerance. C60 was defined as observed plasma concentration at 60 min after administration of enteral feed with 3-OMG. The absorption profile of 3-OMG was used as an indirect measure of gastric emptying function. The analysis was performed on ITT (exposed) Population. Cmax was not analyzed. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles).
Time Frame: At Day 2
Population: ITT (exposed) Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Log (mmol/L)
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
Log (mmol/L)
  C60; Pre-dose | 0.12547 [0.09174 to 0.17159] | 0.12856 [0.09001 to 0.18362]
  C60; post-dose | 0.19960 [0.15935 to 0.25000] | 0.18723 [0.13985 to 0.25065]

24. Secondary Outcome: Derived Tmax of 3-OMG Post Intolerance
Description: Blood samples for PK analysis were collected at Day 2 or Day 3 (or very rarely at Day 4 - only if Day 2 or Day 3 sample could not be obtained) post development of intolerance. Tmax was defined as time to maximum observed plasma concentration of 3-OMG.
Time Frame: At Day 2
Population: PK Population. Data for Tmax was not collected.
Arm/Group | Camicinal 50 mg
Number analyzed (Participants) | 0

25. Secondary Outcome: Percentage of Participants That Became Intolerant
Description: Percentage of participants that became intolerant was calculated. Those participants who developed intolerance were assessed to characterize gastric emptying (GE). Participants who did not develop intolerance were censored at the time of the last available Gastric Residual Volume (GRV) measurement.
Time Frame: Up to Day 7
Population: ITT (exposed) Population. Two participants in the camicinal group and one participant in the placebo group had their last available GRV assessment done prior to first dose and are therefore excluded from this summary.
Measure: Number; unit: Percentage of participants
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 40 | 37
Percentage of participants | 15 | 14

26. Secondary Outcome: Time to Development of Feeding Intolerance
Description: Time required for the development of feeding intolerance was calculated using Kaplan-Meier estimates for time variable. Median and quartiles were not calculable due to the small number of participants developing EN intolerance and mean and standard error of mean were presented.
Time Frame: Up to Day 7
Population: ITT (exposed) Population. Two subjects in the Camicinal group and one subject in the placebo group had their last available GRV assessment done prior to first dose and are therefore excluded from this summary.
Measure: Mean (Standard Error); unit: Hr
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 40 | 37
Hr | 102.9 (5.39) | 108.0 (6.26)

27. Secondary Outcome: GE Assessment as AUC (0-60) Within 24 Hrs of Developing Intolerance and Prior to Change of Treatment Using Acetaminophen
Description: GE assessment within 24 hrs of developing intolerance and prior to change of treatment was analyzed using acetaminophen absorption method. AUC (0-60) was calculated and data was presented for pre-dose Visit (day prior to change of treatment). Geometric mean and 95 percent CI was analyzed.
Time Frame: Day 2
Population: ITT (exposed) Population. Only those participants with data available at pre-dose visit were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: min*ng/mL
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 36
min*ng/mL | 192321.7 [153049.5 to 241671.0] | 222411.3 [161086.4 to 307082.4]

28. Secondary Outcome: GE Assessment as Cmax Within 24 Hrs of Developing Intolerance and Prior to Change of Treatment Using Acetaminophen
Description: GE assessment within 24 hrs of developing intolerance and prior to change of treatment was analyzed using acetaminophen absorption method. Cmax was calculated and data was presented for pre-dose Visit(day prior to change of treatment). Geometric mean and 95 percent CI was analyzed.
Time Frame: Baseline, Day 2, Day 3, Day 4
Population: ITT (exposed) Population. Only those participants with data available at pre-dose visit were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 36
ng/mL | 5482.09 [4529.01 to 6635.72] | 6068.34 [4428.15 to 8316.07]

29. Secondary Outcome: GE Assessment as AUC (0-60) and AUC (0-240) Within 24 Hrs of Developing Intolerance and Prior to Change of Treatment Using 3-OMG
Description: GE assessment within 24 hrs of developing intolerance and prior to change of treatment was analyzed using 3-OMG absorption method. AUC(0-60) and AUC (0-240) was calculated and data was presented for pre-dose Visit (day prior to change of treatment). Geometric mean and 95 percent CI was analyzed.
Time Frame: Baseline, Day 2, Day 3, Day 4
Population: ITT (exposed) Population. Only those participants with data available at pre-dose visit were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: min*mmol/l
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 38 | 34
min*mmol/l
  AUC(0-60); n= 38, 34 | 3.3709 [2.2283 to 5.0993] | 3.8341 [2.5286 to 5.8136]
  AUC(0-240); n= 36, 33 | 31.4065 [23.7921 to 41.4578] | 26.4060 [17.8925 to 38.9703]

30. Secondary Outcome: GE Assessment as C60 Within 24 Hrs of Developing Intolerance and Prior to Change of Treatment Using 3-OMG
Description: GE assessment within 24 hrs of developing intolerance and prior to change of treatment was analyzed using 3-OMG absorption method. C60 was calculated and data was presented for pre-dose Visit (day prior to change of treatment). Geometric mean and 95 percent CI was analyzed.
Time Frame: Baseline, Day 2, Day 3, Day 4
Population: ITT (exposed) Population. Only those participants available at the pre-dose visit were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: mmol/l
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 38 | 34
mmol/l | 0.12547 [0.09174 to 0.17159] | 0.12856 [0.09001 to 0.18362]

31. Secondary Outcome: Number of Participants With Occurrences of Vomiting, Regurgitation and Macroaspiration Episodes
Description: The total number of vomiting, regurgitation and macroaspiration episodes were categorized separately for prior to and post intolerance. Intolerance was considered as start of intolerance treatment. Only the records with non-zero counts were listed.
Time Frame: up to 23 days
Population: Enrolled Population
Measure: Number; unit: Participants
Groups:
- No Treatment: Participant who did not receive treatment.
Arm/Group | Baseline EN Tolerant: Placebo/Camicinal | Baseline EN Tolerant: Camicinal/Metoclopramide | Baseline EN Intolerant: Camicinal | No Treatment
Number analyzed (Participants) | 40 | 44 | 4 | 4
Participants
  Vomiting | 6 | 7 | 0 | 1
  Macroaspiration | 0 | 1 | 1 | 0
  Regurgitation | 1 | 1 | 0 | 0

32. Secondary Outcome: Total GRV for 24 hr Period
Description: Total GRV for each 24 hr period up to 7 days were assessed to determine the effect of GSK962040 vs. Placebo upon the daily GRV. Intolerance was defined as start of the intolerance treatment. The total GRV for each 24hr period was the sum of all available GRV measurements during the period. The 24hr was counted using the same 24hr clock as for the collection of nutritional data.
Time Frame: Up to Day 7
Population: ITT (exposed) Population. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Camicinal 50 mg | Placebo
Number analyzed (Participants) | 42 | 38
mL
  Day 1; n= 36,34 | 37.2 (64.64) | 92.7 (184.83)
  Day 2; n= 34,32 | 118.5 (290.26) | 191.6 (259.93)
  Day 3; n= 29,26 | 169.7 (259.73) | 143.3 (258.46)
  Day 4; n= 23,22 | 131.9 (178.71) | 83.3 (106.55)
  Day 5; n= 19,19 | 185.2 (312.93) | 97.5 (150.45)
  Day 6; n= 15,15 | 180.0 (313.03) | 135.7 (285.43)
  Day 7; n= 12,10 | 85.6 (155.67) | 60.2 (45.66)

33. Secondary Outcome: Log Transformed Derived Plasma Cmax of GSK962040 Prior to Intolerance
Description: Blood samples for PK analysis were collected at Day 2, Day 3, Day 4, Day 7 prior to intolerance. Prior to intolerance was defined as prior to development of intolerance. Cmax was defined as maximum observed plasma concentration of Camicinal. The analysis was performed on PK Population. PK Population comprised of participants in the 'Safety' population for whom a PK sample of Camicinal was obtained and analyzed. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles).
Time Frame: Day 2, Day 3, Day 4, Day 7
Population: PK Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Log (ng/mL)
Arm/Group | Camicinal 50 mg
Number analyzed (Participants) | 42
Log (ng/mL)
  Day 2; n= 25 | 952.55 [740.67 to 1225.04]
  Day 3; n=3 | 748.28 [87.38 to 6408.21]
  Day 4; n= 5 | 1722.74 [1167.35 to 2542.38]
  Day 7; n= 5 | 1206.67 [753.77 to 1931.70]

34. Secondary Outcome: Log Transformed Derived Plasma Cmax of GSK962040 Post Intolerance
Description: Blood samples for PK analysis were collected at Day 2 and Day 4 post development of intolerance. Cmax was defined as maximum observed plasma concentration of Camicinal. The analysis was performed on PK Population. NA indicates that data were not available. SD was not provided if n < 3.
Time Frame: Day 2 and Day 4
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles)
Measure: Geometric Mean (95% Confidence Interval); unit: Log (ng/mL)
Arm/Group | Camicinal 50 mg
Number analyzed (Participants) | 7
Log (ng/mL)
  Intolerance Day 2; n= 2 | 168.56 [NA to NA] — NA indicates that the data were not available.
  Intolerance Day 4; n= 1 | 704.40 [NA to NA] — NA indicates that the data were not available.

35. Secondary Outcome: Derived Tmax of GSK962040 Post Intolerance
Description: Blood samples for PK analysis were collected at Day 2 and Day 4 post development of intolerance. Tmax was defined as time to maximum observed plasma concentration of Camicinal.NA indicates that data were not available. SD was not provided if n<3.
Time Frame: Day 2 and Day 4
Population: as for outcome 34
Measure: Median (Full Range); unit: Hr
Arm/Group | Camicinal 50 mg
Number analyzed (Participants) | 7
Hr
  Intolerance Day 2; n= 2 | 2.717 [1.93 to 3.50]
  Intolerance day 4; n= 1 | 1.500 [1.50 to 1.50]

36. Secondary Outcome: Derived AUC Over the Dosing Period [AUC(0-tau)] of GSK962040 Post Intolerance
Description: Blood samples for PK analysis were collected at Baseline, and at Day 2 and Day 4 post development of intolerance. AUC from time zero extrapolated to infinite time [AUC(0-inf)] was not analyzed.
Time Frame: Day 2 and Day 4
Population: PK Population.
Measure: Geometric Mean (Standard Deviation); unit: min*mmol/l
Arm/Group | Camicinal 50 mg
Number analyzed (Participants) | 1
min*mmol/l
  Intolerance Day 2 | 792.8 (NA) — SD was not provided if n<3
  Intolerance Day 4 | 2698.8 (NA) — SD was not provided if n<3

37. Secondary Outcome: Derived Accumulation Ratio (RO) of GSK962040 Post Intolerance
Description: To estimate the extent of accumulation after repeat dosing, the observed accumulation ratio (Ro) was assessed.
Time Frame: Baseline, Day 2, Day 3, Day 4
Population: PK Population. data were not collected.
Arm/Group | Camicinal 50 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious adverse events (SAEs) were collected for approximately 23 days from start of study treatment until follow up 14 days post last-dose.
Description: AE and SAE analysis was based on Safety Population consisting of all participants who received at least one dose of study treatment.
Arm/Group | Baseline EN Tolerant: Placebo | Baseline EN Tolerant: Camicinal 50 mg | Baseline EN Tolerant: Placebo/Camicinal 50 mg | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg | Baseline EN Intolerant: Camicinal 50 mg | Baseline EN Intolerant: Metoclopramide 10 mg
Serious Adverse Events (participants affected / at risk) | 1/35 | 4/39 | 0/3 | 0/3 | 0/4 | 2/4
Other Adverse Events (participants affected / at risk) | 9/35 | 13/39 | 2/3 | 2/3 | 0/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline EN Tolerant: Placebo (N=35) | Baseline EN Tolerant: Camicinal 50 mg (N=39) | Baseline EN Tolerant: Placebo/Camicinal 50 mg (N=3) | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg (N=3) | Baseline EN Intolerant: Camicinal 50 mg (N=4) | Baseline EN Intolerant: Metoclopramide 10 mg (N=4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline EN Tolerant: Placebo (N=35) | Baseline EN Tolerant: Camicinal 50 mg (N=39) | Baseline EN Tolerant: Placebo/Camicinal 50 mg (N=3) | Baseline EN Tolerant: Camicinal 50 mg/ Metoclopramide 10 mg (N=3) | Baseline EN Intolerant: Camicinal 50 mg (N=4) | Baseline EN Intolerant: Metoclopramide 10 mg (N=4)
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 2 | 3 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin graft failure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Device dislocation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.